## STATISTICAL ANALYSIS PLAN (SAP)

**Study Title**: A Phase 2, Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group, Study to Investigate the Safety and Tolerability of Multiple Dose Administration of CSL112 in Subjects with Moderate Renal Impairment and Acute Myocardial Infarction

**Investigational Medicinal Product**: CSL112

Protocol Number: CSL112\_2001

Version: 1.0 Final

Version Date: 03-AUG-2017

**Sponsor**: CSL Behring

This document includes information and data that contain trade secrets and privileged or confidential information which is the property of CSL Behring LLC and/or its affiliates ("CSL"). This information must not be made public without written permission from CSL. These restrictions on disclosure will apply equally to all future information supplied to you.

**CONFIDENTIAL** 

Template: DAT-SOP-01-T01 Version Number: 1.0

## CSL Behring

Statistical Analysis Plan

Protocol Number: CSL112 2001 Product Name: CSL112

## Signature page

#### **Authors:**

| CSL Behring Study<br>Statistician | PPD | | Date (dd/mmm/yyyy) |
|-----------------------------------|----------|------|--------------------|
| Author: | —<br>PPD | , MS | PPD |

| ESP Lead<br>Statistician | Name | Signature | Date (dd/mmm/yyyy) |
|--------------------------|------|-----------|--------------------|
| Author: | PPD | PPD | PPD |
| Title: | | | |
| Company: | PPD | | |

### **CSL Behring**

Statistical Analysis Plan

Protocol Number: CSL112\_2001 Product Name: CSL112

## Approvers:

By signing below I approve of this version of the Statistical Analysis Plan.

| | Name | Date (dd/mmm/yyyy) |
|--------------|-------------|--------------------|
| Approved by: | PPD | PPD |
| Title: | | |
| Company: | CSL Behring | |


## **Table of Contents**

| Table | of Contents | 4 |
|-------|-------------------------------------------------------|----|
| 1 N | Iodification History | 8 |
| 2 L | ist of Abbreviations | 9 |
| 3 P | urpose | 11 |
| 4 S | tudy Design | 12 |
| 4.1 | Study Design | |
| 4.1.1 | Screening Period | |
| 4.1.2 | Active Treatment Period | |
| 4.1.3 | Safety Follow-Up Period | |
| 4.2 | Objectives and Endpoints | |
| 4.2.1 | Primary Study Hypotheses | 19 |
| 4.3 | Study Treatments. | 19 |
| 4.4 | Schedule of Assessments | 19 |
| 4.5 | Randomization Procedures and Blinding | 19 |
| 4.5.1 | Derived Stratification | 20 |
| 4.6 | Determination of the Sample Size | 20 |
| 4.7 | Planned Interim Analyses and Reviews | 20 |
| 4.7.1 | Interim Analyses Other Than Sample Size Re-estimation | 20 |
| 4.7.2 | Interim Sample Size Re-estimation | 21 |
| 4.7.3 | Data Safety Monitoring Board Reviews | 21 |
| 5 C | hanges in the Conduct of Planned Analyses | 21 |
| 6 S | tudy Analysis Populations | 22 |
| 6.1 | All Subjects Screened [SCR] Population | 22 |
| 6.2 | Intent-to-Treat [ITT] Population | 22 |
| 6.3 | Safety [SAF] Population | 22 |
| 6.4 | Pharmacokinetic [PK] Population. | 22 |
| 6.5 | | 23 |
| 6.6 | | 23 |

## **CSL** Behring

## Statistical Analysis Plan

Protocol Number: CSL112\_2001

| 7 | General Considerations | 23 |
|------|---------------------------------------------------|----|
| 7.1 | Multicenter Studies | 24 |
| 7.2 | Treatment Descriptors | 25 |
| 7.3 | Multiple Comparisons and Multiplicity | 25 |
| 8 | Data Handling Conventions. | 25 |
| 8.1 | Missing Data | 25 |
| 8.1. | 1 Imputation of Non-Date Missing Data | 25 |
| 8.1. | .2 Imputation of Partial Dates | 26 |
| 8.2 | Derived Variables | 28 |
| 8.2. | .1 Reference Dates | 29 |
| 8.2. | .2 Study Day and Relative Day for Safety Measures | 29 |
| 8.2. | .3 Durations | 29 |
| 8.2. | .4 Baseline Definition | 30 |
| 8.2. | .5 Change from Baseline | 30 |
| 8.2. | .6 Multiple Assessments | 30 |
| 8.2. | .7 Actual Treatment | 31 |
| 8.2. | .8 Derived Variables | 31 |
| 8.2. | | 33 |
| 8.3 | Values of Potential Clinical Importance | 33 |
| 8.3. | .1 Laboratory Parameters. | 33 |
| 8.3. | .2 ECG Parameters | 34 |
| 8.3. | 3.3 Vital Signs | 35 |
| 9 | Study Population | 36 |
| 9.1 | Disposition of Subjects | 36 |
| 9.2 | Protocol Deviations | 36 |
| 9.3 | Eligibility Criteria | 38 |
| 9.4 | Demographic and Baseline Characteristics | 38 |
| 9.5 | Concomitant Medications and Procedures | 43 |
| | Efficacy. | |
| 11 | Safety Analyses | 44 |
| 11.1 | 1 Co-primary Endpoints | 44 |

Product Name: CSL112

Protocol Number: CSL112\_2001

| 11.2 Analysis of Co-primary Endpoints | 47 |
|---|---|
| 11.2.1 Sensitivity Analyses of Co-primary endpoints | 48 |
| 11.2.2 Subgroup Analyses of Co-primary Endpoints | 49 |
| 11.3 Extent of Exposure | 49 |
| 11.4 Adverse Events | 50 |
| 11.5 Adverse Events of Special Interest (AESI) | 51 |
| 11.5.1 Stage 3 Acute Kidney Injury | 52 |
| 11.5.2 Drug Hypersensitivity | |
| 11.5.3 Potential Hy's Law Cases | 53 |
| 11.5.4 Hemolysis | 53 |
| 11.5.5 Bleeding Events | 53 |
| 11.6 Deaths and Serious Adverse Events | 53 |
| 11.7 Adverse Events Leading to Discontinuation of Study Study, and Other Significant Adverse Events | |
| 11.8 Adverse Drug Reactions | 55 |
| 11.9 Pregnancies | 56 |
| 11.10 Clinical Laboratory Evaluations | 56 |
| 11.10.1 Hematology, Serum Biochemistry, and Liver Functi | on from the Central Laboratory |
| | 56 |
| 11.10.2 Hepatic Injury Assessment | 59 |
| 11.10.3 Stage 3 Acute Kidney Injury | |
| 11.10.4 Hy's Law | |
| 11.10.5 Hemolysis | |
| 11.10.6 Drug Hypersensitivity | |
| 11.10.7 Local Laboratory Assessments | |
| 11.10.8 Urinalysis | |
| 11.10.9 Evaluation of Immunogenic Potential | |
| 11.11 Other Safety Measures | |
| 11.11.1 Vital Signs | 63 |
| 11.11.2 ECG | 63 |
| 11.11.3 Physical Examination | 64 |
| 11.12 Treatment Compliance | 64 |
| 12 Pharmacokinetic Analyses | 65 |

Product Name: CSL112

## **CSL** Behring

## Statistical Analysis Plan

Protocol Number: CSL112\_2001 Product Name: CSL112

| 12.1 | Measured and Baseline-Corrected Plasma Apolipoprotein A-I and Phosphat Concentrations | - |
|---|---|---|
| 12.2 | Population PK Analysis | 65 |
| 12.3 | Deriving and Summarizing Pharmacokinetic Parameters | 66 |
| 13 C | ···· | 66 |
| 13.1 | CCI | 66 |
| 13.2 | CCI | 67 |
| 13.3 | CCI | 68 |
| 13.4 | CCI | 68 |
| REFI | ERENCES | 69 |
| Appe | endices | 70 |
| 13.5 | List of Tables, Listings, and Figures | 70 |
| 13.6 | List of Preferred Terms within Standardised MedDRA Queries | 78 |
| 13.6. | 1 Co-Primary Endpoint Renal SAEs | 78 |
| 13.6. | 2 Drug Hypersensitivity | 79 |
| 13.6. | 3 Bleeding Events | 87 |
| 13.6. | 4 Hemolysis | 100 |
| 13.7 | Source Data for Identifying Baseline Medications of Interest | 101 |

# 1 Modification History

| Version | Effective Date | Author of<br>Modification | Reason for Change |
|---|---|---|---|
| 0.1 (Draft) | 10NOV2016 | PPD<br>CSL Statisitician | N/A – First Draft Version. |
| 0.2 (Draft) | 26DEC2016 | PPD Statistician | First Draft for Review. |
| 0.3 (Draft) | 03JAN2017 | Statistician | Updates inline with Draft Shell Creation. |
| 1.0 (Draft) | 22FEB2017 | Statistician | Updates based on First Round of CSL Feedback. |
| 1.1 (Draft) | 07MAR2017 | PPD Statistician | Updates based on v1.0 Feedback from CSL Biostatistics. |
| 1.2 (Draft) | 25APR2017 | PPD Statistician | Updates incorporated for production of Dry Run 1. |
| 2.0 (Draft) | 22MAY2017 | PPD Statistician | Updates based on Feedback v.1.1 and the Dry Run 1 from CSL. |
| 2.1 (Draft) | 20JUN2017 | PPD Statistician | Updates incorporated for production of Dry Run 2. |
| 2.2 (Draft) | 19JUL2017 | PPD Statistician | Updates based on Feedback v.2.1 and the Dry Run 2 from CSL. |
| 2.3(Draft) | 03AUG2017 | PPD Statistician | Minor updates in build up to Database Lock. |
| 1.0 (Final) | 03AUG2017 | PPD Statistician | Rounded for Final Versioning and Signatures. |


## 2 List of Abbreviations

| ABCA1 | ATP-Binding Cassette Transporter 1 |
|---------|---------------------------------------------------|
| aCS | Abnormal, Clinically Significant |
| AE | Adverse Event |
| AESI | Adverse Events of Special Interest |
| AKI | Acute Kidney Injury |
| ALT | Alanine Aminotransferase |
| AMI | Acute Myocardial Infarction |
| aNCS | Abnormal, Not Clinically Significant |
| ApoA-I | Apolipoprotein A-I |
| CCI | |
| AST | Aspartate Aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BARC | Bleeding Academic Research Consortium |
| BMI | Body Mass Index |
| BUN | Blood Urea Nitrogen |
| CI | Confidence Interval |
| CKD-EPI | Chronic Kidney Disease Epidemiology Collaboration |
| CSR | Clinical Study Report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CTMS | Clinical Trial Management System |
| CV | Cardiovascular |
| CV % | Coefficient of Variation |
| DBP | Diastolic Blood Pressure |
| DSMB | Data Safety Monitoring Board |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| eGFR | estimated Glomerular Filtration Rate |
| EOS | End of Study |
| FDA | Food and Drug Administration |
| FMC | First Medical Contact |
| Gmean | Geometric Mean |


Statistical Analysis Plan

Protocol Number: CSL112\_2001 Product Name: CSL112

| GSD | Geometric Standard Deviation |
|----------------|------------------------------------------------|
| CCI | |
| CCI | |
| IB | Investigator's Brochure |
| ICH | International Conference on Harmonisation |
| CCI | |
| IND | Investigational New Drug |
| IP | Investigational Product |
| ISO | International Organization for Standardization |
| ITT | Intent-to-Treat |
| IV | Intravenous |
| IRT | Interactive Response Technology |
| KDIGO | Kidney Disease Improving Global Outcomes |
| LDH | Lactate Dehydrogenase |
| CCI | |
| LLN | Lower Limit of Normal |
| LVEF | Left Ventricular Ejection Fraction |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | Myocardial Infarction |
| mRNA | Messenger Ribonucleic Acid |
| n | Number of Observations |
| NCI | National Cancer Institute |
| NOAEL | No Observed Adverse Effect Level |
| NSTEMI | Non-ST Segment Elevation Myocardial Infarction |
| CCI | |
| PC | Phosphatidylcholine |
| PD | Pharmacodynamic |
| PK | Pharmacokinetic |
| PT | Preferred Term |
| QTcB | Bazett's QT correction |
| QTcF | Fridericia's QT correction |
| R <sub>A</sub> | Accumulation Ratio |
| RI | Renal Impairment |


Statistical Analysis Plan

Protocol Number: CSL112\_2001 Product Name: CSL112

| SAE | Serious Adverse Event |
|-------|--------------------------------------------|
| SAF | Safety Population |
| SAP | Statistical Analysis Plan |
| SBP | Systolic Blood Pressure |
| SCR | All Subjects Screened |
| SD | Standard Deviation |
| SI | International System |
| SMQ | Standard MedDRA Query |
| SOC | System Organ Class |
| STEMI | ST Segment Elevation Myocardial Infarction |
| TEAE | Treatment-Emergent Adverse Event |
| TLF | Tables, Listings and Figures |
| ULN | Upper Limit of Normal |
| URS | User Requirements Specification |
| USA | United States of America |
| WBC | White Blood Cells |
| WHODD | World Health Organization Drug Dictionary |

## 3 Purpose

This statistical analysis plan (SAP) provides a detailed and complete description for the final analysis of the study CSL112\_2001 to support the Clinical Study Report (CSR). Mock tables, listings, and figures shells are provided in separate supporting documents.

This SAP complies with the International Conference on Harmonisation (ICH) Harmonised Tripartite Guideline Topic E9, Statistical Principles for Clinical Trials. It is based upon the following study document:

- Study Protocol Amendment 1 (dated 6<sup>th</sup> June 2016)
- Country-specific Clinical Protocol for the United States of America (USA) (dated 6<sup>th</sup> June 2016)

Selected pharmacokinetic (PK) CCI analysis plans will be provided as separate documents.

All decisions regarding the final analysis of the study results, as defined in this SAP document, have been agreed prior to Database Lock of the study data.


### 4 Study Design

### 4.1 Study Design

This is a phase 2, multicenter, double-blind, randomized, placebo-controlled, parallel-group study to assess the safety and tolerability of up to 4 weekly intravenous (IV) administrations of CSL112 6g compared with Placebo in subjects with moderate renal impairment (RI) and acute myocardial infarction (AMI).

The study will consist of a screening period and 2 study periods: an Active Treatment Period during which subjects will receive 4 IV infusions of investigational product (IP) over approximately 22 days and a Safety Follow-up Period, beginning approximately 7 days after the last infusion and lasting approximately 30 days. The Active Treatment Period and the Safety Follow-up Period are defined in Sections 4.1.2 and 4.1.3 respectively. The final analysis to support the CSR will be performed after study completion.

The study will be considered complete when either the pre-specified study completion is reached (all randomized subjects either complete Visit 8/Study Day 60, have withdrawn from the study, or have been lost to follow-up) or the study is terminated early based on the recommendation of the independent Data and Safety Monitoring Board (DSMB) and endorsement by the Steering Committee.

The main study will enroll approximately 81 subjects who will be randomly assigned in a 2:1 ratio to receive infusions of CSL112 6g (54 subjects) versus placebo (27 subjects) to evaluate safety and tolerability. Randomization will be stratified by estimated Glomerular Filtration Rate (eGFR) (30 - <45 mL/min/1.73 m<sup>2</sup> or 45 - <60 mL/min/1.73 m<sup>2</sup>, as calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation [Levey et al, 2009; Stevens et al, 2010]) and by medical history of diabetes requiring current treatment with any anti-diabetic medication (yes or no).

To ensure at least one-third of randomized subjects have eGFR between 30 - <45 mL/min/1.73 m<sup>2</sup>, randomization of subjects with eGFR between 45 - <60 mL/min/1.73 m<sup>2</sup> will be restricted to no more than 54 subjects.




Figure 4-1: Study Overview

AMI = acute myocardial infarction; IV = intravenous; FMC = first medical contact.

The study will consist of screening and 2 study periods: an Active Treatment Period (approximately 29 days) and a Safety Follow-up Period (approximately 30 days from the end of the Active Treatment Period).

Subjects will be assessed for eligibility during screening and up to and including randomization (Visit 1 and Visit 2 before infusion), which may occur no later than 5 days after FMC for the index AMI. Eligible subjects meeting all inclusion criteria and none of the exclusion criteria will receive four 2-hour IV infusions of investigational product (CSL112 6g or Placebo), a minimum of 7 days apart, during an Active Treatment Period lasting approximately 4 weeks.

## 4.1.1 Screening Period

The Screening Period is defined as the period of time leading up to and including randomization and expected to last for approximately 5 days. Randomization must occur within 5 days of first medical contact (FMC) for the index AMI.

Note that at the beginning of the study, sites in the United States were required to ensure that prior to any first infusion, subjects were clinically stable at least 48 hours after the index MI, resulting in a Screening Period of 7 days. However the DSMB made the recommendation to permit earlier administration of the first infusion bringing the Screening Period for sites in the United States inline with sites in the rest of the world (5 Days). Further details are given in Section 5 regarding the DSMB recommendation.


Note that Screening and randomization of subjects may occur on the same day (Study Day 1 of the Active Treatment Period) provided that the minimum time for assessment of renal function stability is adhered to before administration of the first infusion of IP. Refer to Section 8.2.1.2 of the study protocol (Amendment 1, 6<sup>th</sup> June 2016) for further details.

#### 4.1.2 Active Treatment Period

The Active Treatment Period is expected to last for approximately 28 days and begins at the time of a subject's first infusion. The end of the Active Treatment Period occurs at the end of the day of Visit 7 (Study Day 29).

If the Visit 7 assessment was not performed, then the end of the Active Treatment Period is the date of the subject's last administration of study medication + 10 (7+3) calendar days. If an event occurred at any time on the 10<sup>th</sup> day after the day of the last administration, this would be deemed to be within the Active Treatment Period.

## 4.1.3 Safety Follow-Up Period

The Safety Follow-up Period is expected to last for approximately 30 days and will begin the day after the end of the Active Treatment Period. Subjects will return to the study clinic at Visit 8 (Study Day 60) for assessment of adverse events (AEs) and other safety procedures.

## 4.2 Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| The primary objective of this study is to assess the renal safety of CSL112 in subjects with moderate RI and AMI after administration of up to 4 weekly infusions of CSL112. | receive up to 4 weekly administrations of CSL112 will be assessed by co-primary endpoints of the incidences of treatment-emergent |
| | <ul> <li>(1) renal serious adverse events (SAEs) as defined below, and</li> <li>(2) Acute kidney injury (AKI), defined as an absolute increase in serum creatinine (central laboratory) from baseline ≥ 0.3 mg/dL (26.5</li> </ul> |


| Objectives | Endpoints |
|---|---|
| | µmol/L) during the Active Treatment Period that is sustained upon repeat measurement by the central laboratory no earlier than 24 hours after the elevated value. If no repeat value is obtained [due, for example, to loss to follow-up or protocol violation], a single serum creatinine value that is increased from baseline ≥ 0.3 mg/dL (26.5 μmol/L) during the Active Treatment Period would also fulfil the definition of AKI. |
| | Treatment-emergent is defined as occurring at or after the start of the first infusion. |
| | Baseline for determination of AKI is defined as the pre-infusion central laboratory serum creatinine level on Study Day 1 (Visit 2). |
| | A renal SAE is defined as any SAE with a Medical Dictionary for Regulatory Activities (MedDRA) preferred term (PT) included in the Acute Renal Failure narrow Standard MedDRA Query (SMQ) or a PT of Renal Tubular Necrosis, Renal Cortical Necrosis, Renal Necrosis, or Renal Papillary Necrosis. |
| | Incidence rates will be based on the number of subjects with at least 1 occurrence of the event of interest; that is, a subject with 2 treatment-emergent renal SAEs or 2 instances of AKI will be counted once. |
| Secondary | |
| <ol> <li>The secondary objectives of the study are:</li> <li>To further characterize the safety and tolerability of CSL112 in subjects with moderate RI and AMI.</li> <li>To characterize the PK of CSL112 after multiple dose administration in subjects with moderate RI and AMI.</li> </ol> | Secondary safety and tolerability endpoints include: 1. The occurrence of any treatment-emergent adverse event (TEAE) throughout the study. 2. The occurrence of treatment-emergent adverse drug reactions or suspected |


| Objectives | Endpoints |
|---|---|
| | adverse drug reactions defined as: |
| | <ul> <li>a. A TEAE, including local tolerability events, that begin during or within 1 hour of the end of an infusion, or</li> <li>b. A TEAE reported as causally related to the administration of study treatment or which the Sponsor determined to be causally related to the administration of study treatment, or</li> <li>c. A TEAE for which the Investigator's causality assessment is missing or indeterminate, or</li> <li>d. All TEAEs for which the incidence in an active treatment arm exceeds the exposure-adjusted incidence rate in the placebo arm by 30% or more, provided the difference in incidence rates is 1% or more.</li> </ul> |
| | 3. Changes from baseline (ie, pre-infusion on Study Day 1) through to the end of the Active Treatment Period in renal status defined as: |
| | <ul> <li>a. Absolute changes from baseline in serum creatinine as follows:</li> <li>i. ≤ baseline value</li> <li>ii. &gt; 0 to &lt; 0.3 mg/dL</li> <li>iii. ≥ 0.3 to ≤ 0.5 mg/dL</li> <li>iv. &gt; 0.5 mg/dL</li> </ul> |
| | <ul> <li>b. Increases in serum creatinine that are sustained for ≥ 24 hours upon repeat measurement as follows: <ol> <li>i. ≥ 1.5 x baseline values</li> <li>ii. ≥ 2 x baseline value</li> <li>iii. ≥ 3 x baseline value</li> <li>iv. serum creatinine ≥ 4.0 mg/dL (353.6 μmol/L)</li> </ol> </li> </ul> |
| | <ul> <li>c. Initiation of renal replacement therapy</li> <li>d. Decrease in eGFR by ≥ 25% from</li> </ul> |
| | baseline starting during the Active |


| Objectives | Endpoints |
|---|---|
| | Treatment Period and that is sustained at the final study visit |
| | 4. Change from baseline (ie, pre-infusion on Study Day 1) in hepatic status that occurs during the Active Treatment Period and that is sustained for ≥ 24 hours upon repeat measurement as follows: |
| | <ul> <li>a. Alanine Aminotransferase (ALT) &gt; 3 x upper limit of normal (ULN)</li> <li>b. ALT &gt; 5 x ULN</li> <li>c. ALT &gt; 10 x ULN</li> <li>d. Serum total bilirubin &gt; 1.5 x ULN (Note: For subjects with a history of Gilbert's syndrome, this assessment will be based on direct bilirubin.) a</li> <li>e. Serum total bilirubin &gt; 2 x ULN (Note: For subjects with a history of Gilbert's syndrome, this assessment will be based on direct bilirubin.)</li> <li>f. Possible Hy's Law cases, as defined in the Food and Drug Administration (FDA) Guidance for Industry: Drug- Induced Liver Injury: Premarketing Clinical Evaluation (July 2009; see Section 9.1.3.3 of the study protocol for definition of Hy's Law).</li> </ul> |
| | 5. The occurrence of treatment-emergent bleeding events as defined by the Bleeding Academic Research Consortium (BARC) criteria (Mehran et al, 2011) from the start of the first infusion until the end of the Safety Follow-up Period. |
| | 6. Clinically significant changes in clinical laboratory test results (serum biochemistry, hematology, and urinalysis), physical examination findings, body weight, electrocardiograms (ECGs), and vital signs (blood pressure, pulse rate, and body temperature). |


| Objectives | Endpoints |
|---|---|
| | 7. The occurrence of binding antibodies specific to apoA-I and/or CSL112. |
| | Secondary PK Endpoints |
| | Baseline (ie, pre-infusion on Study Day 1)-corrected plasma apoA-I concentrations |
| | Baseline-corrected plasma PC concentrations |
| | 3. Concentration in plasma at End-of-<br>Infusion for apoA-I and PC |
| | 4. Accumulation ratio (R <sub>A</sub> ) for apoA-I and PC |
| CCI | |

<sup>&</sup>lt;sup>a</sup> This is a correction from the original Protocol text, which specified indirect bilirubin was to be used for subjects with a history of Gilbert's Syndrome, see Section 5.


### 4.2.1 Primary Study Hypotheses

There are no statistical hypothesis tests for this study.

### 4.3 Study Treatments

Subjects receive four, 2-hour IV infusions of IP (CSL112 6g or Placebo), 7 to 10 days apart, during a 4-week Active Treatment Period, with all 4 infusions administered within 30 days from Study Day 1 (Visit 2).

#### 4.4 Schedule of Assessments

The schedules of assessments for the study can be found in the synopsis of the study protocol.

## 4.5 Randomization Procedures and Blinding

Eligible subjects were to be randomized in a 2:1 ratio to receive active treatment versus placebo by means of interactive response technology (IRT). Randomization was to be stratified by eGFR (30 to < 45 mL/min/1.73m<sup>2</sup> or 45 to < 60 mL/min/1.73m<sup>2</sup>) and by medical history of diabetes requiring current treatment with any anti-diabetic medication (yes or no). This randomization scheme results in 4 different strata.

- 30 <45 mL/min/1.73 m<sup>2</sup> with medical history of diabetes requiring current treatment with any anti-diabetic medication.
- 30 <45 mL/min/1.73 m<sup>2</sup> without medical history of diabetes requiring current treatment with any anti-diabetic medication.
- 45 <60 mL/min/1.73 m<sup>2</sup> with medical history of diabetes requiring current treatment with any anti-diabetic medication.
- 45 <60 mL/min/1.73 m<sup>2</sup> without medical history of diabetes requiring current treatment with any anti-diabetic medication.


The eGFR values were to be calculated by the IRT using the CKD-EPI equation and local laboratory values at Visit 2 (Study Day 1). The IRT system then assigned the appropriate study treatment to each subject within each stratum.

The IRT used centralized randomization and fixed-size blocks: to ensure the study blind was maintained, a CSL statistician/delegate not directly involved in the analysis of study results was to prepare the study randomization code. The unblinded CSL statistician/delegate was to keep the randomization code on file.

To ensure adequate numbers of randomized subjects with eGFR between 30 - <45 mL/min/1.73 m<sup>2</sup>, randomization of subjects with eGFR between 45 - <60 mL/min/1.73 m<sup>2</sup> was to be restricted to no more than 54 subjects.

#### 4.5.1 **Derived Stratification**

For the purpose of Safety analyses, stratification will be derived based on data as reported within the database. The eGFR values will be calculated using the Visit 2 (Day 1, Before Infusion) serum creatinine values from the Central Laboratory, whilst the medical history of diabetes requiring current treatment with any anti-diabetic medication will be assigned as recorded on the medical history page of the CRF.

No imputation will be performed in the event that a subject has a missing value for the central laboratory serum creatinine.

## 4.6 Determination of the Sample Size

No formal sample size calculations were performed. The sample size for this study was planned to meet regulatory considerations for treatment-emergent renal event characterization; it was not powered for statistical testing of the co-primary endpoints.

With a sample size of 81 (54 CSL112 6g: 27 Placebo), the study will detect (at least one observed occurance) with 80% probability, a treatment-emergent event with a true incidence of 3% in the active group and 2% overall.

## 4.7 Planned Interim Analyses and Reviews

## 4.7.1 Interim Analyses Other Than Sample Size Re-estimation

No formal interim analyses are planned for this study.


### 4.7.2 Interim Sample Size Re-estimation

Sample size re-estimation is not planned for this study.

## 4.7.3 Data Safety Monitoring Board Reviews

An external program-level DSMB will independently evaluate safety data to assess whether a safety signal has emerged that would warrant a change in the conduct of the study. The DSMB will also review all trial data if one or more criteria of the study level stopping rules are met. The role of the DSMB and the data review schedules are described in detail in the protocol and DSMB charter. The DSMB could recommend a change to the protocol to ameliorate any safety concerns, as specified in the program-level DSMB charter.

## 5 Changes in the Conduct of Planned Analyses

Section 2.2.2 of (and then throughout) the protocol incorrectly specifies the use of Indirect Bilirubin as replacement for Total Bilirubin, for subjects with a history of Gilbert's syndrome when assessing Bilirubin related secondary endpoints. This has been correctly amended in this SAP to use Direct Bilirubin.

On 13<sup>th</sup> February 2017 after reviewing the available data of approximately 35% of subjects who had received two infusions of investigational product and had pre-infusion safety data available prior to the third infusion at Visit 5, the DSMB recommended to reduce the minimum time between IV contrast and the first assessment for renal stability and dosing in the United States from 48 hours to at least 12 hours.

For subjects who had not undergone angiography with IV contrast, the first infusion would now occur no earlier than 12 hours after the subject is considered to be clinically stable after the index Myocardial Infarction (MI). As a result of this recommendation, and as per the adaptive language in the country specific USA protocol, the duration of screening was also reduced so that the screening period up to and including randomization must occur within 5 days of FMC for the index MI (reduced from 7 days).

After this recommendation, the duration of screening and the minimum time from IV contrast to first dose (or minimum time from FMC to first dose if angiography not performed) was harmonized globally.


### 6 Study Analysis Populations

### 6.1 All Subjects Screened [SCR] Population

The all subjects screened (SCR) population will consist of all subjects who provided written informed consent to undergo study screening procedures.

## 6.2 Intent-to-Treat [ITT] Population

The Intent-to-Treat (ITT) population will consist of all subjects in the SCR population who were randomized to 1 of the 2 treatment groups. Analyses based on this population will use the treatment to which the subject was randomized and the stratification assigned by the IRT, regardless of the treatment actually received or the true stratum to which a subject belongs. Any subject who is allocated a treatment randomization number will be considered to have been randomized.

## 6.3 Safety [SAF] Population

The Safety (SAF) population will consist of all subjects in the ITT population who receive at least a partial dose of IP. Analyses based on this population will use the actual treatment received and the derived stratum (See Section 4.5.1) to which a subject belongs, regardless of the treatment and stratum assigned by the IRT.

In cases where a subject receives both CSL112 6g and Placebo, the actual treatment received will be considered to be CSL112 6g.

The SAF population will be used in the analysis of all safety endpoints, including the coprimary endpoints.

## 6.4 Pharmacokinetic [PK] Population

The PK population will consist of all subjects in the SAF population who have at least one measurable plasma concentration of apoA-I or PC.

For displays based on the PK population, subjects will be classified according to actual treatment received and the derived stratum (See Section 4.5.1) to which they belong.




#### 7 General Considerations

Analysis datasets will be created according to the Clinical Data Interchange Standards Consortium (CDISC) standards, and data will be displayed according to reporting standards in this SAP and the tables, listings and figures (TLF) shells.

SAS version 9.4 or higher will be used to perform all data analyses and to generate the TLFs.

Continuous variables will be summarized in terms of the number of observations (n), mean, standard deviation (SD), median, 25<sup>th</sup> percentile, 75<sup>th</sup> percentile, minimum, and maximum. Additional descriptive statistics (eg, the coefficient of variation) may be reported when appropriate.

Categorical variables will be summarized using frequency counts and percentages. Analyses that use other descriptive statistics will have the specific descriptive statistics required identified with the analysis in the applicable SAP section.

All listings will include subject number and treatment group. The laboratory normal reference ranges will be provided and clinical laboratory test results outside the normal reference range will be flagged as abnormal in the laboratory data listings.

Summary statistics of central tendency will be reported to one more decimal place than the collected data. Summary statistics of variability will be reported to one more decimal place than the commensurate measure of central tendency. For example, the


mean and median for age will be reported to one decimal place because it is collected in whole years. The SD of age will then be reported to 2 decimal places. Descriptive percentages and proportions will be displayed to one decimal place. Durations for AEs, will be displayed to the nearest integer.

Formatting for dates and times will follow the International Organization for Standardization (ISO) 8601 format:

- Dates only yyyy-mm-dd
- Times only hh:mm or hh:mm.ss
- Dates and times yyyy-mm-ddThh:mm or yyyy-mm-ddThh:mm:ss

In general, for by-visit summaries, data recorded will be presented for the nominal visit. Unscheduled measurements will not be included in by-visit summaries, but will be eligible to contribute to the End of Study (EOS) value, will be included in the determination of best/worst case values (eg, shift tables) and will appear in listings.

Subjects who discontinue IP prematurely, having signed informed consent, will be followed for AEs as specified in the protocol and complete early termination procedures, which are the same as those conducted at Visit 7 (Day 29). Subjects who have discontinued IP early should continue to be followed for safety through Visit 8 (Day 60).

Listings will include scheduled, unscheduled, retest and early discontinuation data where recorded.

Any deviations from the analyses in this SAP will be identified in the CSR.

#### 7.1 Multicenter Studies

The study is planned to be conducted at approximately 38 sites in the United States, Germany, Hungary, the Netherlands and Israel. Some exploratory subgroup analyses will be performed by country. Data from all participating sites will be pooled prior to analysis.

A summary of enrolment by site will be produced.


## 7.2 Treatment Descriptors

The treatment descriptors are "CSL112 6g" and "Placebo".

## 7.3 Multiple Comparisons and Multiplicity

No statistical hypothesis testing will be performed in this study, therefore no adjustments for multiplicity will be made.

## 8 Data Handling Conventions

Treatment assignments will be applied to the clinical data at the time of the Database Lock based on the randomization schedule, which will be merged using the Randomization Number obtained from the eCRF to obtain the correct treatment assignment.

## 8.1 Missing Data

Missing data occurs when any requested data are not provided, leading to blank fields on the electronic case report form (eCRF). These data will be indicated by the use of a "blank" in subject listing displays. Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data.

## 8.1.1 Imputation of Non-Date Missing Data

Data from assessments that are not conducted because a subject withdrew from the study at any time or permanently discontinued study treatment, before completing all infusions, will not be considered missing data and no imputation for such values will be done.

Subjects with the designation of treatment relationship for AEs and SAEs missing will have the worst case assumed to impute the relationship; ie, if the investigator's assessement of relationship to study treatment is missing it will be assumed to be "Yes". There will be no other imputation for missing data other than as described in Section 8.1.2 for partial dates and times.


In the event that the study is terminated early, all available data will be listed and a review carried out by the study team to assess which statistical analyses are to be performed.

## 8.1.2 Imputation of Partial Dates

Imputed dates are used for slotting events to the appropriate study time periods and for sorting in data listings and will not be used to derive relative day, duration (eg, duration of AEs), or elapsed time variables and as a result will not displayed in any listings.

Partial date imputation will follow ADaM conventions. The ADaM approach is to populate the numeric date variables with the imputed date and add a flag variable to the dataset that indicates the level of imputation.

The flag variable can contain the values: blank, 'D', 'M', 'Y'.

- blank: indicates that no imputation was done
- D = 'Day': indicates that the day portion of the date is imputed
- M = 'Month': indicates that the month and day portions of the date are imputed
- Y = 'Year': indicates that the entire date (year, month, and day) is imputed

Algorithms for imputing partial dates for AEs and medications are below.

#### **Adverse Events**

If an AE start or end date is either completely or partially missing, then the duration of the AE will be set to missing.

| Date | Missing Element(s) | Rule |
|---|---|---|
| Start Date | Day, Month, and Year | Do not impute completely missing AE start dates. |
| | | → The AE will be deemed treatment emergent if the AE end date does not indicate that the AE ended prior to the study treatment start date. |
| | Day and Month. | <ul> <li>If the study treatment start date is not missing: <ul> <li>→ If the year of the AE start date is the same as the year of study treatment start date then</li> <li>■ If the AE end date indicates the AE ended prior to the study treatment start date then set the AE start date to January 1.</li> <li>■ Otherwise set the AE start date to the study treatment start date.</li> </ul> </li> </ul> |
| | | Otherwise set the AE start date to January 1. |


| Date | Missing Element(s) | Rule |
|---|---|---|
| | Day Only | <ul> <li>If the study treatment start date is not missing: <ul> <li>→ If the month and year of the AE start date are the same as the month and year of study treatment start date then</li> <li>■ If the AE end date indicates the AE ended prior to the study treatment start date then the AE start date to the 1st of the month.</li> <li>■ Otherwise set the AE start date to the study treatment start date.</li> </ul> </li> <li>● Otherwise set the AE start date to the 1st of the month.</li> </ul> |
| End Date | Day, Month, and Year | No imputation for completely missing AE end dates; as applicable, report the AE as ongoing and the AE duration as missing. |
| | Any Partial Date | No imputation for partial AE end dates; as applicable report the date as recorded and the AE duration as missing. |

#### **Concomitant Medications:**

Imputations in the concomitant medication dataset will be performed for start and end dates as necessary to derive the prior/concomitant nature of the medication. Imputed dates will be recorded in the concomitant medication analysis dataset with a flag variable as previously described to indicate the level of imputation. The start and end dates will be used to classify medications as taken prior, during, and/or after study treatment.

| Date | Missing Element | Rule |
|---|---|---|
| Start Date | Day, Month, and Year | • Do not impute completely missing medication start dates; all values that depend on this date will be set to missing. |
| | | → The medication will be deemed to be a prior<br>medication if the medication end date indicates<br>that the medication could not have started after<br>study treatment start. |
| | | → Otherwise the medication will be deemed to be concomitant. |
| | Day and Month | If the study treatment start date is not missing: → If the year of the medication start date is the same as the year of the study treatment start date then If the medication end date indicates the medication ended prior to the study treatment start date then set the medication start date to January 1. Otherwise set the medication start date to the study treatment start date. |
| | | Otherwise set the concomitant medication start date to January 1. |


| Date | <b>Missing Element</b> | Rule |
|---|---|---|
| | Day Only | If the study treatment start date is not missing: → If the month and year of the medication start date is the same as the month and year of the study treatment start date then |
| End Date | Day, Month and Year | Do not impute completely missing medication end dates; all values that depend on this date will be set to missing. → The medication will be deemed to be concomitant and ongoing. |
| | Day and Month | <ul> <li>If the medication partial end date contains the year only, set the medication end date to the earliest of [December 31, or the date of the last completed Safety assessment visit including subject completion, date of withdrawal from the study, date of loss to follow-up].</li> <li>If the partial medication end date contains the month and year, set the medication end date to the earliest of [the last day of the end month reported, the date of the last completed Safety assessment, date of withdrawal from the study or date of loss to follow-up].</li> </ul> |
| | Day Only | |

If the start or end dates of a medication is recorded as "unknown" these will be treated as missing for the purposes of assigning as prior or concomitant.

### 8.2 Derived Variables

The following sections provide a general description of the derived and transformed variables to be used in data analyses. Separate analysis dataset specifications provide full details on all data derivations and transformations.


#### 8.2.1 Reference Dates

The safety reference date is defined as the date of the first infusion of study treatment. This safety reference date will be used to assign study periods relative to study treatment.

### 8.2.2 Study Day and Relative Day for Safety Measures

Data presentations by visit, will use scheduled visits. For example, Visit 7 is targeted to occur at scheduled Study Day 29 but due to the visit window, may occur at Relative Day 31. It should be noted that Relative Day is distinct from Study Day, and that there is no Relative Day 0.

Relative Day will be calculated from the start of first infusion (time zero [0 h] on Study Day 1) as;

If the date of the assessment/event is on or after the date of start of first infusion then:

• Relative Day = (date of assessment/event - date of start of first infusion) + 1.

If the date of the assessment/event is prior to the date of start of first infusion then:

• Relative Day = (date of assessment/event – date of start of first infusion).

Relative Day will be used to show start/stop day of assessments and events, and will appear in every listing where an assessment date or event date appears.

In the situation where the assessment/event date is partial or missing, Relative Day, and any corresponding durations will appear missing in the listings.

#### 8.2.3 **Durations**

Durations of events (eg, the duration of an AE or a medication) will be calculated in days using the following formula:

• (End Date – Start Date) + 1.

Durations calculated in days will use dates only.

Duration of infusions will be calculated in hours (h) using the following formula:


• (End Date/Time – Start Date/Time).

Other durations in the study will be presented (eg, ECG parameters); however, as these values come directly from raw data and no calculation is required, these are not detailed in this document.

#### 8.2.4 Baseline Definition

Baseline for both laboratory and non-laboratory data is defined as the most recent preinfusion, non-missing value prior to or on the date of first study treatment infusion.

## 8.2.5 Change from Baseline

Change from baseline will only be calculated for measures that have post-baseline records.

Change from baseline for safety measures will be calculated as:

Visit value – Baseline value.

Percentage change from baseline will be calculated as:

• ((Change from baseline) / Baseline value) \* 100

If either the baseline or visit value are missing, then the change from baseline and percentage change from baseline will also be set to missing.

## 8.2.6 Multiple Assessments

All data will be reported according to the nominal visit date for which it was reported (that is, no visit windows will be applied during dataset creation).

Unscheduled serum creatinine assessments form a critical part of the co-primary endpoint for AKI identification. After an initial elevation ( $\geq 0.3 \text{ mg/dL}$ ) is observed, an unscheduled repeat measurement should occur no earlier than 24 hours after the initial elevation. See Section 11.1 for the details of the programming algorithm for identification and confirmation of events.

All unscheduled data will be included in worst case post-baseline summaries.


Data from all assessments (scheduled and unscheduled), including multiple assessments, will be included in listings.

### 8.2.7 Actual Treatment

The subjects' actual treatment will be assigned from the "End of Study (Unblinded Data File)" as a data extract from the IRT. The external vendor, Cenduit, will provide this file to Quintiles after confirmation of Database Lock. Reconciliation of kit numbers and materials dispensed/infused was conducted within the IRT. Further details on the contents of this file are provided in Section 10.3 of the User Requirements Specification (URS) v9.0 dated 8<sup>th</sup> March 2017.

In the event that a subject receives a study treatment that is different from the assigned treatment, then assigning the actual treatment received will follow this rule:

• CSL112 6g overrides Placebo

For example, if a subject had 3 doses of Placebo and a single dose of CSL112 6g, then the actual treatment assignment would be CSL112 6g.

#### 8.2.8 Derived Variables

#### Derivation of Body Mass Index (BMI)

BMI will be calculated using the following formula:

BMI 
$$(kg/m^2)$$
 = Weight  $(kg) / [Height (m)]^2$ 

Using the height measured at Screening and the weight measured at Day 1 (if available). If weight at Day 1 is not available, the assessment at Screening will be used (if available). If neither is available, then BMI is missing.

#### Derivation of Direct Bilirubin (Local)

The calculation of Direct Bilirubin is only applicable when both Total Bilirubin and Indirect Bilirubin are given in the raw local laboratory data. No calculation of Indirect Bilirubin is required.

Direct Bilirubin ( $\mu$ mol/L) = Total Bilirubin ( $\mu$ mol/L) - Indirect Bilirubin ( $\mu$ mol/L)


## Derivation of eGFR

For the purpose of safety analysis, the eGFR value will be recalculated using the Visit 2 (Day 1, Before Infusion) serum creatinine values from the Central Laboratory for eGFR (Central) and the Local Laboratory for eGFR (Local) using the CKD-EPI equations in Table 1:

**Table 1: CKD-EPI Equations** 

| Race and Sex Serum Creatinine mg/dL (µmol/L) | | Equation |
|---|---|---|
| Black | | |
| Female | ≤ 0.7 (≤ 62) | eGFR = 166 * (SeCr/0.7) <sup>-0.329</sup> * 0.993 <sup>Age</sup> |
| | > 0.7 (> 62) | eGFR = 166 * (SeCr/0.7) <sup>-1.209</sup> * 0.993 <sup>Age</sup> |
| Male | ≤ 0.9 (≤ 80) | eGFR = 163 * (SeCr/0.9) <sup>-0.411</sup> * 0.993 <sup>Age</sup> |
| | > 0.9 (>80) | eGFR = 163 * (SeCr/0.9) <sup>-1.209</sup> * 0.993 <sup>Age</sup> |
| White or Other | | |
| Female | ≤ 0.7 (≤ 62) | eGFR = 144 * (SeCr/0.7) <sup>-0.329</sup> * 0.993 <sup>Age</sup> |
| | > 0.7 (> 62) | eGFR = 144 * (SeCr/0.7) <sup>-1.209</sup> * 0.993 <sup>Age</sup> |
| Male | ≤ 0.9 (≤ 80) | eGFR = 141 * (SeCr/0.9) <sup>-0.411</sup> * 0.993 <sup>Age</sup> |
| | > 0.9 (> 80) | eGFR = 141 * (SeCr/0.9) <sup>-1.209</sup> * 0.993 <sup>Age</sup> |

The CKD-EPI equation can be expressed as a single equation:

• eGFR =  $141 \times \min(\text{SeCr/}\kappa, 1)^{\alpha} \times \max(\text{SeCr/}\kappa, 1)^{-1.209} \times 0.993^{\text{Age}} \times 1.018$  [if female]  $\times 1.159$  [if black],

where SeCr is serum creatinine,  $\kappa$  is 0.7 for females and 0.9 for males,  $\alpha$  is -0.329 for females and -0.411 for males, min indicates the minimum of SeCr/ $\kappa$  or 1, and max indicates the maximum of SeCr/ $\kappa$  or 1. In Table 1: the multiplication factors for race and sex are incorporated into the intercept, which results in the different intercepts for age and sex combinations.

Derived eGFR values will be presented to two decimal places.


### 8.2.9 Study Time Periods for Other Medications

Medications, other than study treatment, will be designated as "Prior" and/or "Concomitant" based on start and end dates relative to first dose of study treatment. For instances where the medication date is either partial or missing, refer to Section 8.1.2.

Designate as "Prior" if the medication start date is prior to study treatment start date; if subject has not taken any study treatment; or the medication start date is missing.

Designate as "Concomitant" if the medication start date is before the study treatment end date and the medication end date is either after the study treatment start date or missing.

Note that a medication may be both "Prior" and "Concomitant, ie, the categories are not mutually exclusive.

Baseline medications are defined as any medication that started on or prior to the date of first infusion, and the end date is either after the date of first infusion or missing (implying the medication is ongoing).

Prior to Index MI medications are defined as those medications that either ended or were ongoing 1 day prior to the date of the subjects Index MI event.

## 8.3 Values of Potential Clinical Importance

## 8.3.1 Laboratory Parameters

A laboratory value that is outside the reference range can be categorized as either a high abnormal value (a value above the ULN) or low abnormal value (a value below the lower limit of the normal (LLN)). A laboratory parameter can take on both high and low abnormal values at different Safety assessment visits. Note that an abnormal laboratory value is not necessarily one of potential clinical interest.

Increases in specific laboratory values associated with the secondary endpoints are:

- Absolute changes from baseline in serum creatinine:
  - $\rightarrow \leq$  Baseline value
  - $\rightarrow$  > 0 to <0.3 mg/dL
  - $\rightarrow$   $\geq 0.3$  to  $\leq 0.5$  mg/dL †
  - $\rightarrow$  > 0.5 mg/dL †
- † Potential clinical significance.


• Increases in serum creatinine sustained for  $\geq 24$  hours upon repeat measurement:

- $\rightarrow \geq 1.5$ x baseline value,
- $\rightarrow$  > 2.0x baseline value.
- $\rightarrow$  > 3.0x baseline value
- $\rightarrow \geq 4.0 \text{ mg/dL} (353.6 \,\mu\text{mol/L})$

An additional summary will be presented for single instances of increases in serum creatinine, i.e. without assessment of whether those increases were sustained.

- A decrease in eGFR (Central)  $\geq 25\%$  from baseline starting during the Active Treatment Period and that is sustained at the final study visit
- Changes from baseline in hepatic status that occur during the Active Treatment Period and that are sustained for  $\geq 24$  hours upon repeat measurement as follows:
  - $\rightarrow$  ALT > 3x ULN,
  - $\rightarrow$  ALT > 5x ULN,
  - $\rightarrow$  ALT > 10x ULN
  - $\rightarrow$  Serum Total Bilirubin † > 1.5x ULN,
  - $\rightarrow$  Serum Total Bilirubin † > 2x ULN

An additional summary will be presented for single instances of increases, i.e. without assessment of whether those increases were sustained.

† Note that for subjects with a history of Gilbert's syndrome, serum bilirubin assessments will be based on direct bilirubin. The calculation of direct bilirubin for local laboratory values is given in Section 8.2.8.

Secondary endpoints as specified in the protocol section 2.2 include clinically significant changes in clinical laboratory test results (serum biochemistry, hematology, and urinalysis) with Grade 3 and 4 Laboratory Abnormalities, as potentially clinically significant laboratory test results, see Table 9:.

#### 8.3.2 ECG Parameters

Abnormal quantitative ECG measurements will be identified in accordance with the predefined markedly abnormal criteria in Table 2:.


Table 2: Markedly Abnormal Quantitative ECG Measurements

| ECG parameter | Markedly Abnormal Change |
|---|---|
| | >450 msec |
| | >480 msec |
| QT uncorrected,<br>QTcB and QTcF | >500 msec |
| | >30 msec increase from baseline |
| | >60 msec increase from baseline |
| Heart rate | ≥ 120 bpm during active treatment and an increase of ≥15 bpm from baseline |
| | ≤ 50 bpm during treatment and a decrease of ≥15 bpm from baseline |
| DD/OD interval | <120 msec during treatment and a normal baseline value |
| PR/QR interval | >210 msec during treatment and a normal baseline value |
| QRS >110 msec during treatment and a normal baseline value | |

# 8.3.3 Vital Signs

Markedly abnormal quantitative Vital Signs measurements will be identified in accordance with the predefined markedly abnormal criteria detailed in Table 3: in Section 8.3.3.

Table 3: Vital Signs Markedly Abnormal Criteria

| Variable | Unit | Low | High |
|---|---|---|---|
| Systolic Blood | mmHg | ≤ 90 AND a decrease from | ≥ 180 AND an increase from |
| Pressure | mining | baseline ≥ 20 | baseline ≥ 20 |
| Diastolic Blood | mmHg | ≤ 50 AND a decrease from | ≥ 105 AND an increase from |
| Pressure | mining | baseline ≥ 15 | baseline ≥ 15 |
| Pulse | bpm | ≤ 50 AND a decrease from | ≥ 120 AND an increase from |
| | | baseline ≥15 | baseline ≥ 15 |
| Body Temperature | °C | NA | $\geq$ 38.3 °C AND an increase |
| Body Temperature | | | from baseline $\geq 1.1$ |
| Weight | kg | Percentage decrease from | Percentage increase from |
| weight | | baseline ≥ 7.0 % | baseline ≥ 7.0 % |


## 9 Study Population

## 9.1 Disposition of Subjects

Summary tables with columns identified by IP group: (CSL112 6g, Placebo, Total) will be produced for the following;

- Total number of subjects in each of the analysis populations described in Section
   6.
- Total number of subjects in each of the 4 randomization strata: eGFR 30 <45 mL/min/1.73 m<sup>2</sup> or 45 <60 mL/min/1.73 m<sup>2</sup> and by medical history of diabetes requiring current treatment with any anti-diabetic medication (yes or no).
- Study treatment status, including subjects who completed the study (defined as all subjects who completed Visit 8 (Day 60)), discontinued IP (including reasons for discontinuation), or withdrew consent for the study.
- Subject completion by visit.
- Subjects screened, (including screen failures) and subjects randomized to IP.
- Duration of Follow-up, ie, the time from randomization to last contact.

Reasons for study withdrawal and study treatment discontinuation will be presented in the order they are displayed in the eCRF.

The following details will be provided in listings:

- Screen failure subjects, including reason for screening failure.
- Reasons for study withdrawal including the date of withdrawal.
- Reasons for study treatment discontinuation. The listing will include last dose date, cumulative dose, and reasons for study treatment discontinuation.
- Reasons for discontinuation of IP and withdrawal of consent from the study will be listed for each such subject.
- Differences between actual treatment received and randomized, as well as between strata allocation based on central laboratory values (derived) and the randomized assignment.

#### 9.2 Protocol Deviations

All instances of deviations from the protocol will be documented in the Clinical Trial Management System (CTMS) log. A deviation occurs when an investigator site, or study subject, does not adhere to protocol stipulated requirements. Deviations will be assessed by CSL as they are reported and categorized as either Major or Minor.

Both Major and Minor protocol deviations for subjects in the ITT population will be summarized, displaying the number and percentage of subjects with any protocol deviation as well as the categories for the deviations. All protocol deviations will be listed.

Refer to the Protocol Deviation Management Plan (v1.0 dated November 1<sup>st</sup> 2016) for complete details on the handling of protocol deviations.

A further by subject listing will be prepared for deviations related to infusion durations. The following deviations will be identified programmatically:

- Infusion duration < 2 hours and the infusion rate exceeds 3 mg/kg/min of sucrose
- Infusion duration > 3 hours and
  - $\rightarrow$  < 80% volume of IP was administered, or
  - $\rightarrow$  > 120% volume of IP was administered.

CCI

 $\mathsf{CC}$ 

CCI

Additional by subject listings will be produced for subjects who:

- Received IP different to their randomized treatment
- Were randomized but did not meet eligibility criteria
- Were allocated to the incorrect stratum in IRT based on the eGFR (Local) value.
- Were allocated to the incorrect stratum in IRT based on the Medical History data for Diabetes Mellitus.

The eGFR (Local) value will be calculated using the local laboratory baseline serum creatinine, age, sex, and race. For the derivation of eGFR see Section 8.2.8.

- eGFR (Local)
  - $\rightarrow$  < 30 mL/min/1.73 m<sup>2</sup>
  - $\rightarrow$  30 < 45 mL/min/1.73 m<sup>2</sup>
  - $\rightarrow$  45 <60 mL/min/1.73 m<sup>2</sup>
  - $\rightarrow \geq 60 \text{ mL/min/1.73 m}^2$


### 9.3 Eligibility Criteria

A summary of Inclusion/Exclusion criterion failed for screen failures in addition to a by subject listing will be produced. As subjects may fail to meet more than one Inclusion and/or Exclusion criterion, the percentages across criteria may not sum to 100%.

### 9.4 Demographic and Baseline Characteristics

The following demographic data will be summarized by treatment group:

• Age (years)  $\rightarrow$  18 to < 65,  $\rightarrow$  ≥ 65 to < 75,  $\rightarrow$  ≥ 75 to < 85,  $\rightarrow$  > 85

In addition to summarization as a categorical variable, age (years) will also be summarized as a continuous variable.

- Sex
- Ethnicity
- Race

For subjects reporting more than one Race category, classify as "Racial Combination" group.

• Country

The following baseline characteristics will be summarized by treatment group for the ITT population.

- Height (cm)
- Weight (kg)
- BMI (kg/m<sup>2</sup>) (See Section 8.2.8)
- eGFR from IRT using Local Laboratory data from Visit 2 (or Screening).
  - $\rightarrow$  30 < 45 mL/min/1.73 m<sup>2</sup>
  - $\rightarrow$  45 < 60 mL/min/1.73 m<sup>2</sup>

The eGFR (IRT) value will be calculated by the IRT from the serum creatinine obtained by the local laboratory at Visit 2, or Screening if the screening visit and randomization occur on the same day.


Statistical Analysis Plan

Protocol Number: CSL112\_2001 Product Name: CSL112

- eGFR (Central)
  - $\rightarrow$  < 30 mL/min/1.73 m<sup>2</sup>
  - $\rightarrow$  30 < 45 mL/min/1.73 m<sup>2</sup>
  - $\rightarrow$  45 <60 mL/min/1.73 m<sup>2</sup>
  - $\rightarrow > 60 \text{ mL/min/1.73 m}^2$

The eGFR (Central) value will be calculated using the central laboratory baseline serum creatinine, age, sex, and race. For the derivation of eGFR see Section 8.2.8.

The eGFR (Central) values will be summarized both categorically using these groupings and as a continuous variable using univariate statistics. A summary of the agreement between randomized and derived strata allocation will be produced.

- Disease characteristics at screening.
  - $\rightarrow$  Type of Index MI
    - ST Segment Elevation Myocardial Infarction (STEMI)
    - Non-ST Segment Elevation Myocardial Infarction (NSTEMI)

The following targeted medical history will be summarized by treatment group for the ITT population.

- Prior MI
- Stable angina
- Unstable angina
- Coronary revascularization or surgery (prior to Index MI)
- Congestive heart failure
- Peripheral artery disease
- Clinically significant valvular heart disease
- Clinically significant heart rhythm disorder
- Cerebrovascular disease
- Clinically significant bleeds
- Hypertension
- Gilbert's Syndrome
- Chronic kidney disease
- Dyslipidemia or use of treatment for dyslipidemia
- Diabetes mellitus
- Smoking/tobacco use

All other medical history within 3 months before the screening visit is entered into the eCRF as free text and will be coded using MedDRA version 20.0 and summarized by treatment group, System Organ Classes (SOC) and PT. By subject listings for all medical history data will also be produced.


Statistical Analysis Plan

Protocol Number: CSL112\_2001 Product Name: CSL112

- Baseline Medications of Interest
  - → Aspirin
  - → Anti-thrombotics
  - → Anti-platelets
  - → Beta blockers,
  - → Angiotensin-Converting-Enzyme Inhibitor (ACE-I) or Angiotensin Receptor Blockers (ARB).
  - → Anti-hyperlipidemic Consisting of statins and other lipid modifying agents.

For the timing rules regarding identification of medications being taken at baseline, refer to Section 8.2.9. An external source dataset (Excel format) containing the full set of individual medications of interest will be provided by CSL.

- Baseline Statin Use
  - → High dose/intensity
  - → Moderate dose/intensity
  - → Low dose/intensity
  - $\rightarrow$  None

Table 5: contains the anatomical therapeutic chemical (ATC) and World Health Organization drug dictionary (WHODD) codes in addition to the dose thresholds for identifying the moderate and high dose/intensity statins (Stone NJ, et al, 2014).


Table 5: Identification of Moderate and High Dose/Intensity Statins

| | | ATC I1 4 | | Daily Dose T | hreshold |
|---|---|---|---|---|---|
| Preferred Name | WHODD Code | ATC Level 4<br>Code | ATC Level 4 Text | Moderate<br>Intensity | High<br>Intensity |
| ATORVASTATIN | 1326101001 | | | | |
| LIPITOR | 1326102016 | C10AA | HMG COA<br>REDUCTASE | ≥10 to <40 mg | ≥ 40mg |
| ATORVASTATIN<br>CALCIUM | 1326102001 | 0.101.11 | INHIBITORS | | <u> </u> |
| ROSUVASTATIN | 1588601001 | | | | |
| CRESTOR | 1588602002 | C10AA | HMG COA<br>REDUCTASE | ≥5 to <20 mg | ≥ 20mg |
| ROSUVASTATIN<br>CALCIUM | 1588602001 | 010111 | INHIBITORS | _5 to 20 mg | ≥ 2011ig |
| SIMVASTATIN | 848101001 | C10AA | HMG COA<br>REDUCTASE<br>INHIBITORS | ≥20 to <80 mg | ≥ 80mg |
| ZOCOR | 00848101004 | C10AA | HMG COA<br>REDUCTASE<br>INHIBITORS | | ≥ 80mg |
| PRAVASTATIN | 880401001 | G10.4.4 | HMG COA | > 40 | |
| LOVASTATIN | 896701001 | C10AA | REDUCTASE<br>INHIBITORS | ≥ 40mg | |
| FLUVASTATIN | 1224501001 | | HMG COA | | |
| FLUVASTATIN<br>XL | 1224502107 | C10AA | REDUCTASE<br>INHIBITORS | ≥ 80 mg | |
| PITAVASTATIN | 6470001001 | C10AA | HMG COA<br>REDUCTASE<br>INHIBITORS | ≥ 2 mg | |
| INEGY (ezetimibe and simvastatin) | 1726001001 | | | | |
| VYTORIN<br>(ezetimibe and<br>simvastatin) | 1726001002 | C10BA | HMG COA REDUCTASE INHIBITORS IN COMBINATION WITH | | ≥ 10mg and<br>≥ 40mg, |
| EZETIMIBE<br>W/SIMVASTATIN | 1726001003 | | OTHER LIPID<br>MODIFYING AGENTS | respective | |
| EZETIMIBE<br>/SIMVASTATIN | 1726001029 | | | | |


Statistical Analysis Plan

Protocol Number: CSL112\_2001 Product Name: CSL112

Subjects with simultaneous use of the medications in Table 6: will be considered to be on a high dose/intensity statin. Use of either drug at these levels without the other does not constitute high dose/intensity statin use.

Table 6: Identification of Combination High Dose/Intensity Statins

| D. C. LV | WHODD C. I | Daily Dose Threshold High Intensity |
|---|---|---|
| Preferred Name | WHODD Code | |
| EZETIMIBE and SIMVASTATIN | 01587001001<br>00848101001 | |
| EZETIMIBE and ZOCOR | 01587001001<br>00848101004 | |
| ZETIA and SIMVASTATIN | 01587001003<br>00848101001 | > 10 |
| ZETIA and ZOCOR | 01587001003<br>00848101004 | $\geq 10$ mg and $\geq 40$ mg, respectively |
| EZETROL and SIMVASTATIN | 01587001002<br>00848101001 | |
| EZETROL and ZOCOR | 01587001002<br>00848101004 | |

Summary statistics on the following timing durations, overall and by country will also be presented:

- Index MI to Angiography
- Angiography to Randomization
- Angiography to First Infusion
- Randomization to First Infusion
- Index MI to First Infusion
- Angiography to Local Laboratory Sample used to Determine Eligibility

The following listings will be provided:

- Demographic characteristics
- Race
- Pregnancy testing
- Follicle Simulating Hormone (FSH) testing
- Targeted and non-targeted medical history
- Medications of Interest


- Medications of Interest taken the day prior to Index MI,
- Medications of Interest taken after Index MI and continuing at Randomization.
- Use of renal replacement therapy

Renal replacement therapy will be identified using the MedDRA terms in Table 7: and must begin after the start of the first infusion and no later than the end of the Active Treatment Period.

**Table 7: Qualifying Renal Replacement Therapies** 

| MedDRA Preferred Term Code | MedDRA Preferred Term |
|----------------------------|-------------------------------|
| 10061105 | Dialysis |
| 10034660 | Peritoneal dialysis |
| 10018875 | Haemodialysis |
| 10066338 | Continuous haemodiafiltration |
| 10038533 | Renal transplant |

### 9.5 Concomitant Medications and Procedures

Medications will be coded using the WHODD (1st March 2017 Enhanced Version). They will be summarized in alphabetical order of generic term and grouped by the ATC code. Procedures will be coded using MedDRA version 20.0 and will be summarized in alphabetical order of PT. The summaries of medications and procedures will show the number and percentage of subjects taking the medications/receiving the procedures.

Listings based on the ITT population will also be provided.

Medications other than study treatment, and procedures will be designated as "Prior" and/or "Concomitant" based on the start and end dates relative to first dose of study treatment as described in Section 8.2.9.

Note that a medication may be designated as both "Prior" and "Concomitant, ie the categories are not mutually exclusive.

Prohibited medication use will be monitored by the CSL medical monitoring team via regular review of the medication data. If any prohibited medications are discovered they will be entered into the CTMS protocol deviation log, under the deviation category of "Concomitant Medication Criteria".

Individual summaries of both prior and concomitant medications and procedures will be produced. Subjects with multiple instances of the same medication/procedure will be counted only once in each designation of prior or concomitant.


### 10 Efficacy

No efficacy analyses will be performed.

### 11 Safety Analyses

All safety analyses will be based on the SAF as defined in Section 6.

### 11.1 Co-primary Endpoints

The renal safety profile of CSL112 in subjects with moderate RI and AMI who receive up to 4 weekly administrations of CSL112 6g will be assessed by co-primary endpoints of the incidences of:

- Treatment-emergent renal SAEs,
- Treatment-emergent AKI

Incidence rates will be based on the number of subjects with at least 1 occurrence of the event of interest; that is, a subject with 2 treatment-emergent renal SAEs or 2 instances of AKI will be counted once for the respective co-primary endpoint.

Note that treatment emergent renal SAEs can occur at any time on or after the first infusion, whilst AKI events must occur within the Active Treatment Period.

#### **Renal Serious Adverse Events**

Treatment-emergent is defined as occurring anytime on or after the start of the first infusion through to the end of the study.

A renal SAE is defined as any SAE with a MedDRA PT included in the following;

- Acute Renal Failure narrow SMQ (See Section 13.6.1)
- Renal Tubular Necrosis
- Renal Cortical Necrosis
- Renal Necrosis
- Renal Papillary Necrosis


Any renal SAE reported between the start of the first infusion and a subject's final study visit will be a co-primary endpoint event.

Non-serious AEs with any of the above MedDRA PTs do not form part of the Co-Primary Endpoint.

### **Acute Kidney Injury**

Baseline for determination of AKI is defined as the pre-infusion central laboratory serum creatinine level on Study Day 1.

AKI is defined as an absolute increase in serum creatinine from baseline  $\geq 0.3$  mg/dL (26.5 µmol/L) during the Active Treatment Period (See Section 4.1.2.) that is sustained upon repeat measurement by the central laboratory no earlier than 24 hours after the elevated value. If no repeat value is obtained during the Active Treatment Period (eg, due to loss to follow-up or a protocol violation), a single serum creatinine value that is increased from baseline  $\geq 0.3$  mg/dL (26.5 µmol/L) during the Active Treatment Period would also fulfil the definition of AKI.

To identify a subject with an AKI event the following logic will be applied. Note that any given subject may have more than one AKI event during the Active Treatment Period:

- 1. Calculate the change from baseline (mg/dL) for each post-baseline serum creatinine value (including unscheduled assessments) during the Active Treatment Period.
- 2. Order the change values from the earliest to the latest by date and time.
- 3. Evaluating from the earliest to the latest visit, identify the initial increase from baseline of  $\geq 0.3$  mg/dL.
  - a. If the following change from baseline value is also  $\geq 0.3$  mg/dL, and is at least 24 hours after the date and time of the initial increase, then the subject is confirmed to have an AKI event.
  - b. If the following change from baseline value is < 0.3 mg/dL and is at least 24 hours after the initial increase, then this is not an AKI event.
  - c. If the following change from baseline value is < 24 hours after the initial increase, this value should be discounted and the next value in the ordered sequence assessed.


d. If no repeat value at least 24 hours after the initial increase (within the Active Treatment Period) is obtained, then this single increase would also fulfil the definition of AKI.

The end date of the identified AKI event will be determined using the following algorithm for each subject with at least one AKI event:

- 1. Evaluating from the first confirmed increase, determine if there are 2 consecutive change from baseline values < 0.15 mg/dL (ie, with no interspersed changes ≥ 0.15 mg/dL), each at least 24 hours from the preceding change from baseline value.
- 2. If there are 2 consecutive change from baseline values that are < 0.15 mg/dL at least 24 hours apart, then the end date of the AKI event is the date and time of the first increase of these 2 consecutive change from baseline values < 0.15 mg/dL.
- 3. If the subject does not have 2 consecutive change from baseline values that are < 0.15 mg/dL after a confirmed increase, then the end date of the AKI event is missing.

After identifying the first AKI event for a subject and assessing its end date, the algorithms will then be applied to the remaining serum creatinine change values following the initial AKI event to identify any further instances of AKI events for a given subject.

If a subsequent AKI event occurs, and is within 48 hours of the previous event ending, then this will be designated as one single event. This will be determined as follows;

- 1. If the start date and time of the subsequent AKI event is at least 48 hours after the end date and time of the previous AKI event, then the subject is confirmed to have a further instance of an AKI event.
- 2. If the start date and time of the subsequent AKI event is within 48 hours of the end date and time of the previous AKI event, then this is deemed to be the same event.
  - a. The end date and time of the original AKI event will then be replaced with the end date and time of the subsequent AKI event, provided there are no further AKI events within 48 hours of its end date and time. No changes are required to the start date and time of the original AKI event.


### 11.2 Analysis of Co-primary Endpoints

Analysis of the co-primary endpoints will take place at study completion (when all randomized subjects either complete Visit 8/Study Day 60, have withdrawn from the study, or have been lost to follow-up) or after the study is terminated early based on recommendation of the independent DSMB and endorsement by the Steering Committee).

For each co-primary endpoint, a Newcombe-Wilson two-sided 95% confidence interval around the difference in incidence rates will be calculated if at least one event occurs. Otherwise, an exact, one-sided, upper 97.5% confidence interval will be reported for the incidence rate in each treatment arm.

The following will be produced:

- Summaries of the co-primary analysis results. The point estimates of the differences in incidence rates between treatment arms will be provided for each co-primary endpoint separately, along with the Newcombe-Wilson two-sided 95% confidence intervals when at least one event occurs, or otherwise if no event occurs, with the exact, one-sided, upper 97.5% confidence intervals for the incidence rates in each of the treatment arms.
- A summary including the number of AKI events per subject and subject counts for the following day intervals for the duration of AKI events.
  - $\rightarrow 1-7$
  - $\rightarrow$  8-14
  - → 15-21
  - $\rightarrow$  22-28
- A summary of co-primary Renal SAE PTs including the breakdown of information as adjudicated by the CEC.
- A listing of creatinine values for subjects with any AKI events.
- A listing of all AKI events including subject ID, treatment group, change from baseline (mg/dL) in serum creatinine, start date, end date, and duration.
- A listing of all AEs for subjects with any renal SAE.
- Box plots by visit, showing actual and change from baseline values in serum creatinine, as well as eGFR (Central).


• Individual subject series plots of the change from baseline in both central and local laboratory serum creatinine over time, for subjects with at least one central laboratory change from baseline ≥ 0.3mg/dL.

### 11.2.1 Sensitivity Analyses of Co-primary endpoints

A sensitivity analysis of the co-primary endpoints will use independently adjudicated results for the treatment-emergent renal SAE component and local laboratory data for the treatment-emergent AKI component. The same methods as for the primary study analysis described in Section 11.2 will be used.

A further two sensitivity analyses will be performed, the first will include all absolute increases in serum creatinine from baseline  $\geq 0.3$  mg/dL (26.5  $\mu$ mol/L) during the Active Treatment regardless of confirmation. That is the initial increase of 0.3 mg/dL will be enough to qualify as an event for analysis. The same methods as for the primary study analysis described in Section 11.2 will be used.

The second of these sensitivity analyses will repeat the primary analyses, whilst excluding increases in serum creatinine from baseline  $\geq 0.3$  mg/dL (26.5  $\mu$ mol/L) that had a missing confirmatory assessment. That is any increase that was identified as a primary endpoint due to no repeat value being obtained, will be excluded from this sensitivity analysis.

In a separate sensitivity analysis, AKI rates will be compared among subjects whose dosing eligibility was determined in part based on serum creatinine determinations performed 12 to 24 hours after radiographic contrast exposure versus those performed 48± 6 hours after radiographic contrast exposure.

In the event that there are insufficient observations to perform this analysis, (defined as fewer than 15 subjects observed within each timing group) then comparison of the AKI rates among subjects whose dosing eligibility was determined in part based on serum creatinine determinations performed 12 to 48 hours after radiographic contrast exposure versus those performed > 48 hours will be explored.

For either analysis, the difference in placebo-corrected rates between the 2 time-period subgroups will be calculated, along with a 2-sided adjusted Wald 95% confidence interval (Price, Bonett, 2004).

#### **Timing of Serum Creatinine Determinations Algorithm**


The following is the algorithm for calculating the time between contrast and the local laboratory sample used for determining eligibility, which will be used in the sensitivity analysis:

- Timing (hours) = Scr Date/Time (Con Date/Time) where;
  - → Scr is the Sample Collection Date/Time, as reported on the LOCAL1 (or LOCAL4 if Visit 1 and Visit 2 were combined) page of the eCRF, for the Serum Creatinine Value, and
  - → Con is the Date and Time Contrast was Given, as reported on the INDEXMI page of the eCRF.

### 11.2.2 Subgroup Analyses of Co-primary Endpoints

Summaries of co-primary endpoint events and of renal SAEs and AKI events separately will be produced by treatment group for:

- Subjects with eGFR (Central) of <30 mL/min/1.73 m<sup>2</sup>
- Subjects with eGFR (Central) of 30 <45 mL/min/1.73 m<sup>2</sup>
- Subjects with eGFR (Central) of 45 <60 mL/min/1.73 m<sup>2</sup>
- Subjects with eGFR (Central) of >60 mL/min/1.73 m<sup>2</sup>
- Subjects with medical history of diabetes requiring current treatment with any anti-diabetic medication
- Subjects without medical history of diabetes requiring current treatment with any anti-diabetic medication.

The differences in incidence rates between treatment arms will not be provided for the subgroup summaries.

## 11.3 Extent of Exposure

Exposure to IP will be presented for the SAF by treatment group, by infusion and overall. The following will be summarized as well as listed, by treatment group:

- Number of infusions administered per subject
- Number of infusions completed per subject
- Locale for IP Administration

In addition to the above, the following items will be summarized for the by infusion summaries;


Statistical Analysis Plan

Protocol Number: CSL112\_2001 Product Name: CSL112

- Duration of infusions (minutes)
- Number of days between infusions
- Actual volume infused (mL)
- Number of interruptions per infusion

By-subject listings will include, in addition to tabulated data, details regarding infusion modifications, interruptions and any overdoses.

### 11.4 Adverse Events

Adverse Events will be coded using the MedDRA central coding dictionary, Version 20.0 and graded in accordance to the National Cancer Institure (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0. If an event has a missing CTCAE grade, the AE will be assumed to have a grade of 3 for reporting purposes.

All summaries of AEs will include all treatment-emergent AEs (TEAEs), defined as AEs reported at or after the start of the first infusion and presented by SOC and PT. Subjects who have more than one AE recorded for the same PT will only be counted once within that PT. Subjects with multiple PTs will contribute to each PT summary but only once in the overall SOC row.

Summaries of TEAEs will count the number of subjects, not the number of events, that is, subjects with multiple occurrences of the same TEAE will be counted only once.

An overview summary of TEAEs will be produced, including counts and percentages of subjects as well as the number of events, with any:

- TEAE
- Study treatment related TEAE
- Study procedure related TEAE
- Serious TEAE
- Study treatment related serious TEAE
- Fatal TEAE
- Study treatment related fatal TEAE
- TEAE with CTCAE Grade  $\geq 3$
- Line items for TEAEs of special interest identified by PTs (See Section 11.5)
  - → Bleeding Events


- → Potential Hemolysis as Identified Using the Haemolytic Disorders SMO
- → Drug Hypersensitivity Reactions
- Suspected adverse drug reaction (See Section 11.8)
- TEAE leading to study withdrawal
- TEAE leading to permanent discontinuation of study treatment;
- TEAE leading to dose delays
- TEAE leading to dose interruptions
- TEAE leading to skipped doses

The frequency and percentage of TEAEs for each line item of the overview summary will be summarized in descending order of incidence in the CSL112 6g treatment group by PT only. Selected line items will be summarized by SOC and PT.

Missing relationship to study treatment will be imputed as described in Section 8.1.1.

The following summaries will be provided in support of the information described above for TEAEs:

- TEAEs by PT and Maximum Grade
- TEAEs by PT for subgroups based on eGFR (Central) value at the time of randomization.
- TEAEs by PT for subgroups based on diabetic status at the time of randomization

All AEs, regardless of when they were reported, will be listed. Listings will include Subject ID, Derived Stratification Group SOC, Preferred and Verbatim Terms, Relative Start, End and Duration, Severity Grade, SAE (yes or no), Relationship to Treatment, Relationship to Procedure, Any Action Taken and the Outcome of the AE.

The following listings will be provided:

- AEs
- AEs of CTCAE Grade 3 or Higher
- AEs by Treatment showing Subjects Experiencing each PT
- AEs Among Subjects who were Screened but not Treated

## 11.5 Adverse Events of Special Interest (AESI)

The following types of AEs are of special interest for which monitoring and/or expedited reporting by the Investigator is required:


Statistical Analysis Plan

Protocol Number: CSL112\_2001 Product Name: CSL112

- Stage 3 AKI
- Drug hypersensitivity
- Potential Hy's Law cases
- Hemolysis
- Bleeding events

To identify AESI of drug hypersensitivity, hemolysis and bleeding events in the database, a comprehensive list of MedDRA terms based on SMQs will be used to identify the PTs of interest. These are provided in Section 13.6.1.

Summaries by PTs for each of the AESI will be provided separately and consist of;

- AESI Overview for Drug Hypersensitivity Reaction
- Drug Hypersensitivity Reactions by PT
- AESI Overview for Hemolysis
- Hemolysis by PT
- AESI Overview for Bleeding Events as Reported by Investigators
- AESI Overview for Bleeding Events as Adjudicated by the CEC
- Bleeding Events as Reported by Investigators by PT

The following by subject listings will be provided:

- AESI Drug Hypersensitivity Reactions
- AESI Hemolysis
- AESI Bleeding Events

## 11.5.1 Stage 3 Acute Kidney Injury

Acute kidney injury for this purpose is defined as an elevation in serum creatinine during the Active Treatment Period to  $\geq 3x$  the baseline value or a serum creatinine of  $\geq 4.0$  mg/dL (353.6  $\mu$ mol/L, Kidney Disease Improving Global Outcomes [KDIGO] March 2012) that is confirmed by repeat assessment using the central laboratory data.

No identification of Stage 3 AKI will be performed using PTs reported by the investigator, see Section 11.10.3 for further details.

## 11.5.2 Drug Hypersensitivity

If a drug hypersensitivity reaction is suspected, it should be reported as an AE by the investigator. The list of PTs for identifying these drug hypersensitivity reactions are given in Section 13.6.2.


### 11.5.3 Potential Hy's Law Cases

Potential Hy's Law cases for the purpose of AESI identification will be defined as any elevation in ALT > 3x ULN with a concomitant increase in total bilirubin that is > 2x ULN that is confirmed by repeat assessment using the central laboratory data. Aspartate aminotransferase (AST) is not being used in this definition since there may be increases in AST that are due to the index MI event.

No identification of potential Hy's Law will be performed using PTs reported by the investigator, see Section 11.10.4 for further details.

### 11.5.4 Hemolysis

Potential hemolysis will be defined as a decrease in hemoglobin during the Active Treatment Period  $\geq 2$  g/dL from baseline using central laboratory data. See Section 11.10.5 for further details.

In addition, in order to rule out decreases in hemoglobin due to overt blood loss, the Haemolytic disorders SMQ (given in Section 0) will be used to identify hemolysis.

There will be separate summaries for events identified by these two methods.

### 11.5.5 Bleeding Events

Bleeding events will be assessed according to the BARC definition for bleeding events and will be independently adjudicated.

The list of PTs for identifying bleeding events of interest are given in Section 13.6.3.

### 11.6 Deaths and Serious Adverse Events

Adverse events leading to death are recorded on the AE page of the eCRF with an outcome of 'Fatal'. A tabular summary will be prepared displaying the number and percentage of subjects with a fatal AE and primary cause of death (disease under study, SAE related to study treatment, or other).

If there are no deaths on study, then this display will be produced with the text "No deaths reported". Deaths, if any, will also be listed. A supportive listing will be generated to provide subject-specific details on subjects who died.


If there are any deaths, the following summaries will be provided based on the number and percentage of subjects experiencing each unique PT:

- Fatal TEAEs by PT
- Fatal Study Treatment-Related TEAEs by PT

SAEs will be summarized based on the number and percentage of subjects experiencing each unique PT. The following summaries will be provided:

- Treatment-emergent SAEs by PT
- Study treatment-related treatment-emergent SAEs PT

The following listings to support the summaries described above will be provided:

- SAEs
- Fatal AEs
- Deaths Among Subjects who were Screened but not Treated

# 11.7 Adverse Events Leading to Discontinuation of Study Treatment, Withdrawal from the Study, and Other Significant Adverse Events

The following categories of treatment-emergent AEs will be summarized based on the number and percentage of subjects experiencing each unique PT:

- TEAEs Leading to Withdrawal from the Study, by PT
- TEAEs Leading to Permanent Discontinuation of Study Treatment, by PT
- TEAEs Leading to Infusion Delays, by PT
- TEAEs Leading to Infusion Interruptions, by PT
- TEAEs Leading to Skipped Infusions, by PT

The following listings to support the summaries described above will be provided:

- AEs Leading to Withdrawal from the Study
- AEs Leading to Permanent Discontinuation of Study Treatment
- AEs Leading to Infusion Delays
- AEs Leading to Infusion Interruptions
- AEs Leading to Skipped Infusions


### 11.8 Adverse Drug Reactions

An adverse drug reaction (or suspected adverse drug reaction) is defined as either:

- a. A TEAE, including local tolerability events, that begin during or within 1 hour of the end of an infusion, or
- b. A TEAE reported as causally related to the administration of study treatment, or which the sponsor determined to be causally related to the administration of study treatment, or
- c. A TEAE for which the investigator's causality assessment is missing or indeterminate, or
- d. All TEAEs for which the incidence in an active treatment arm exceeds the exposure-adjusted incidence rate in the placebo arm by 30% or more, provided the difference in incidence rates is 1% or more.

A summary of all suspected adverse drug reactions by SOC and PT will be provided along with a supportive by subject listing.

### **Exposure Adjusted Algorithm**

For each PT recorded on the AE page of the CRF, the following algorithm will be applied to define whether or not the PT in question is an adverse drug reaction according to criterion d.

Incidence Rate (IR) =  $\frac{Total\ Number\ of\ Subjects\ with\ Events}{Total\ Number\ of\ Subjects}$  Exposure Adjusted IR  $\frac{Total\ Number\ of\ Subjects\ with\ Events}{Total\ Number\ of\ Subjects\ with\ Events}$ 

 $(EAIR) = \frac{1}{Total\ Number\ of\ Infusions\ Administered\ Across\ All\ Subjects}$ 

Therefore the PT will be considered an adverse drug reaction according to criterion d if and only if both of the following are true;

- Active IR-Placebo IR  $\geq 1\%$ .
- $\left(\frac{Active\ EAIR-Placebo\ EAIR}{Placebo\ EAIR}\times 100\right) \ge 30\%$ , where Placebo EAIR > 0.

If the number of events within the placebo group is 0 (ie, Placebo EAIR = 0), then the PT will be considered to be an adverse drug reaction if (Active IR-Placebo IR)  $\geq 1\%$ .

For adverse drug reactions identified according to criterion d, all subjects experiencing that particular PT will be included in the summary and listing.


### 11.9 Pregnancies

While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or elective termination of a pregnancy for medical reasons will be recorded as an AE or SAE as described in the protocol. If any subject or subject's partner becomes pregnant while on the study, the information will be included in the narratives and no separate table or listing will be produced.

### 11.10 Clinical Laboratory Evaluations

Summaries for worst observations will include data from scheduled and unscheduled visits obtained from the central laboratory data. Other tabular summaries will only include data from scheduled visits obtained from central laboratory data, whilst listings will be prepared for both Central and Local laboratory data along with laboratory specific normal ranges.

For all summaries of clinical laboratory evaluations that reference a baseline value, the definition for the baseline assessment is in Section 8.2.4.

The denominator in any percentage calculations at each scheduled visit will be based on the number of subjects with a non-missing value at the respective visit.

Separate summary tables for hematology, chemistry, liver function, and urinalysis will be produced.

# 11.10.1Hematology, Serum Biochemistry, and Liver Function from the Central Laboratory

The following parameters from the central laboratory will be summarized with descriptive statistics, by treatment group, and scheduled visit. All presentations will use International System (SI) Units.

| Hematology | Serum Biochemistry | Liver Function |
|------------|--------------------|----------------|
|------------|--------------------|----------------|


Statistical Analysis Plan

Protocol Number: CSL112\_2001 Product Name: CSL112

| Hemoglobin | • Albumin | <ul> <li>Alkaline phosphatase</li> </ul> |
|---|---|---|
| Hematocrit | <ul> <li>Total Protein</li> </ul> | • ALT |
| RBC Count and Indices | <ul> <li>Creatinine</li> </ul> | • AST |
| WBC Count, Total and | • eGFR (Central) | <ul> <li>Total Bilirubin</li> </ul> |
| Differentials | Blood Urea Nitrogen | <ul> <li>Direct Bilirubin</li> </ul> |
| → Basophils, | (BUN) | <ul> <li>Indirect Bilirubin</li> </ul> |
| → Eosinophils, | • Urate | |
| → Lymphocytes, | <ul> <li>Glucose</li> </ul> | |
| → Monocytes, | • Calcium | |
| → Neutrophils | <ul> <li>Chloride</li> </ul> | |
| Platelet Count | • Sodium | |
| | <ul> <li>Potassium</li> </ul> | |
| | • Bicarbonate | |

Creatinine is collected using mg/dL, conversion to SI unit of  $\mu$ mol/L is required by multiplying using a factor of 88.4.

Glucose is collected using mg/dL, conversion to SI unit of mmol/L is required by multiplying using a factor of 18.018.

Quantitative laboratory measurements reported as "< X", ie, below the lower limit of normal (BLN), or "> X", ie, above the ULN, will be converted to X for the purpose of quantitative summaries, but will be presented as recorded, ie, as "< X" or "> X" in the listings.

Quantitative laboratory measurements will be compared with the relevant laboratory reference ranges in SI units and categorized as:

- Low: Below the lower limit of the laboratory reference range.
- Normal: Within the laboratory reference range (upper and lower limit included).
- High: Above the upper limit of the laboratory reference range.

The following summaries will be provided for laboratory data by treatment group:

- Actual and change from baseline by visit (for quantitative measurements)
- Shifts from baseline to worst observation in the Active Treatment Period according to normal range criteria (for quantitative measurements and


categorical measurements). The definition of "worst" is detailed in Table 8: for each parameter.

If a subject has a decrease to below the normal range and an increase to above the normal range during the same time interval, then the subject is counted in both the decrease to below the normal range and increase to above the normal range categories.

**Table 8: Definition of Worst Observation by Parameter** 

| Low | Low or High | High |
|------------|-------------|----------------------|
| Hemoglobin | Glucose | Alkaline Phosphatase |
| | | ALT |
| | | AST |
| | | Total Bilirubin |
| | | Direct Bilirubin |
| | | Urine Protein |

By-subject listings of subjects with results outside of the normal range in the Active Treatment Period will also be produced.

For the hepatic and renal laboratory parameters, namely ALT, total bilirubin, serum creatinine, and eGFR (Central) values for the change from baseline at each visit and by treatment group will be presented visually using box plots.

Grade 3 and 4 laboratory abnormalities defined in Table 9: will be designated as clinically significant. These will be summarized by time point and listed.

**Table 9: Grade 3 and 4 Laboratory Abnormalities** 

| <b>Laboratory Parameter</b> | Grade 3 | Grade 4 |
|-----------------------------|---------------|-----------|
| Alkaline phosphatase | > 5 - 20x ULN | > 20x ULN |
| ALT | > 5 - 20x ULN | > 20x ULN |


| <b>Laboratory Parameter</b> | Grade 3 | Grade 4 |
|---|---|---|
| AST | > 5 -20x ULN | > 20x ULN |
| Total bilirubin | > 3x - 10x ULN | > 10x ULN |
| Direct bilirubin | > 3x - 10x ULN | > 10x ULN |
| Creatinine | > 3x Baseline | > 6x ULN |
| Creatinine | > 3 - 6x ULN | > 0X OLIN |
| Glucose | > 250 - 500 mg/dL | > 500 mg/dL |
| Hemoglobin | < 8 g/dL | N/A |
| eGFR | 15 - < 30 mL/min/1.73m <sup>2</sup> | < 15 mL/min/1.73 m <sup>2</sup> |

The proportion of subjects who have missing serum creatinine results will be presented by visit and treatment group and for all subjects.

Individual subject series plots will be provided for all subjects who experience at least one instance of a central laboratory serum creatinine change from baseline  $\geq 0.3 \text{mg/dL}$ .

### 11.10.2 Hepatic Injury Assessment

If any subject has elevation in ALT > 3x ULN with a concomitant elevation in total bilirubin > 2x ULN OR an elevation in ALT > 5x ULN, blood samples should be obtained and sent to the central laboratory within 48 to 72 hours for further testing.

These parameters will be identified in the Central Laboratory data panel using the visit label (VISIT) of "Hepatic Injury Assessment". These unscheduled results will be included in the identification of "worst case" values and a listing of all results will be provided.

# 11.10.3 Stage 3 Acute Kidney Injury

Acute kidney injury for this purpose is defined as an elevation in serum creatinine during the Active Treatment Period to  $\geq 3x$  the baseline value or a serum creatinine of  $\geq 4.0$  mg/dL (353.6  $\mu$ mol/L, Kidney Disease Improving Global Outcomes [KDIGO] March 2012) that is confirmed by repeat assessment using the central laboratory data.

## 11.10.4Hy's Law

Hy's Law as defined in the Guidance for Industry: Drug-induced Liver Injury: Premarketing Clinical Evaluation (2009) is an elevation in AST or ALT > 3x ULN


with a concomitant increase in total bilirubin that is > 2x ULN without initial findings of cholestasis (elevated alkaline phosphatase, defined as > 2x ULN), and with no other reason found to explain the combination of these increased AST/ALT and total bilirubin findings.

Note that the AESI of Potential Hy's Law cases uses a definition that excludes AST values. For further details see Section 11.5.3.

A summary table for the concomitant elevations identified using the Central Laboratory data will be produced. Supportive by subject listings will display the Liver Function parameters from both Central and Local Laboratory data panels for subjects contributing to the summary table.

### 11.10.5 Hemolysis

If a post-infusion hemoglobin value is  $\geq 2$  g/dL below the baseline value and is not explained by overt blood loss, assessment for hemolysis should be performed by the central laboratory. The following parameters will be collected for suspected hemolysis, these data will be listed only. These unscheduled assessments will be included in the identification of any worst case values.

- Hemoglobin Level (Repeated)
- Total, Direct Bilirubin and Indirect Bilirubin (Calculated)
- Serum Haptoglobin
- Lactate Dehydrogenase (LDH)
- Urine Hemosiderin

## 11.10.6 Drug Hypersensitivity

If a drug hypersensitivity reaction is suspected, blood samples should be obtained and sent to the central laboratory for calculation of:

- Quantitative immunoglobulins (IgG, IgA, IgM, IgE)
  - → If IgA is low or not detectable, then anti-IgA antibodies will be assayed
- Complete blood count with differential

These data will be listed only.


### 11.10.7 Local Laboratory Assessments

The local laboratory is to be used for all laboratory tests that must be reviewed in real time such as for study eligibility and dosing decisions. All laboratory test samples also go to the central laboratory for analysis.

Local laboratory data will be presented in the same format as for central laboratory results as well as being listed.

### 11.10.8 Urinalysis

To summarize the categorical results at baseline versus the maximum value observed during the Active Treatment Period, shift tables will be produced for the following parameters reported in the central laboratory data:

- Protein
- Occult Blood (Hemoglobin)

A further summary will be prepared displaying descriptive statistics of the following parameters in addition to those detailed above:

• Specific Gravity  

$$\rightarrow \ge 1.000 - < 1.010$$
  
 $\rightarrow \ge 1.010 - < 1.020$   
 $\rightarrow \ge 1.020$ 

• pH  

$$\rightarrow$$
 < 5.0  
 $\rightarrow$  ≥ 5.0 - < 6.0  
 $\rightarrow$  ≥ 6.0 - < 7.0  
 $\rightarrow$  ≥ 7.0 < 8.0  
 $\rightarrow$  > 8.0

- Bilirubin
- Glucose
- Ketones
- Leukocyte Esterase
- Nitrites
- Urine Erythrocytes
- Urine Leukocytes


All parameters collected from microscopic examination of the sediment (casts, crystals, bacteria, renal tubular epithelial cells, and white blood cells [WBCs]) will be listed only.

Note that screening urinalysis will be locally performed by urine dipstick. Only if dipstick analysis demonstrates high grade proteinuria defined as  $\geq$  3+ (ie,  $\geq$  300 mg/dL), will a urine sample be sent to the central laboratory for urinalysis with microscopy. Hence it is expected that the counts for screening be lower than post screening visits in any summaries.



# 11.10.9 Evaluation of Immunogenic Potential

Immunogenicity testing for serum antibodies to CSL112 and/or apoA-I was performed as a tiered assay suite comprised of screening, confirmatory and titering assays.

A sample with a signal below the cut point in the screening assay was considered negative and a reciprocal titer of 10 was reported.

Any sample with signal above the screening cut point was considered potentially positive and was to be analyzed further using the confirmatory assay.

The confirmatory assay was to follow the same protocol as the screening assay, with the exception of CSL112 being added to detection reagents to demonstrate specificity of signal. If the percent inhibition was below the confirmatory cut point the sample was considered negative and a reciprocal titer of 11 was reported. If a sample had a percent inhibition above the confirmatory cut point it was considered positive and was further tested in the titration assay following an appropriate dilution series. The highest dilution at which the sample result was above the cut point was reported as the reciprocal titer for that sample.


Changes from baseline for these reciprocal titers for serum antibodies to CSL112 and to apoA-I will be summarized by treatment group and a by subject listing provided.

### 11.11 Other Safety Measures

The denominator in percentage calculation at each scheduled visit will be based on the number of subjects with non-missing value at each particular visit.

### 11.11.1 Vital Signs

The following Vital Signs measurements will be reported for this study:

- Systolic Blood Pressure (SBP) (mmHg)
- Diastolic Blood Pressure (DBP) (mmHg)
- Pulse (bpm)
- Temperature (<sup>0</sup>C)
- Weight (kg)

Markedly abnormal quantitative Vital Signs measurements will be identified in accordance with Table 3:. The following summaries will be provided:

- Actual and change from baseline by visit
- Incidence of treatment emergent markedly abnormal vital signs
- Listing of all Vital Signs data and of subjects meeting markedly abnormal criteria

For SBP, DBP and pulse, the change from baseline at each visit and by treatment group will be presented visually using box plots.

### 11.11.2ECG

The following ECG parameters will be reported for this study:

- Pulse (bpm)
- PQ/PR Duration (msec)
- RR Interval (msec)
- QRS Duration (msec)
- QT Interval (msec)


- Overall assessment of ECG (Investigator's judgment):
  - → Normal
  - → Abnormal, Not Clinically Significant (aNCS)
  - → Abnormal, Clinically Significant (aCS)

Corrected QT intervals will be derived and reported using the following formulae:

• Bazett's QT correction (QTcB) Interval (msec)

$$QTcB (msec) = \frac{QT (msec)}{\sqrt{RR (sec)}}$$

• Fridericia's QT correction (QTcF) Interval (msec)

$$QTcF (msec) = \frac{QT (msec)}{\sqrt[3]{RR (sec)}}$$

Markedly abnormal quantitative ECG measurements will be identified according to Table 2:. The following summaries will be provided:

- Actual and change from baseline by visit (for quantitative measurements), including the derived QTcB and QTcF values
- Incidence of treatment emergent markedly abnormal ECG intervals
- Shift from baseline to last assessment during Active Treatment Period according to overall assessment (for both quantitative and categorical measurements)
- Listing of all ECG data and of subjects meeting markedly abnormal criteria

### 11.11.3 Physical Examination

Any abnormal physical examination findings considered by the Investigator as clinically significant at the time of screening will be documented as Medical History. Any clinically significant changes occurring between screening and the end of the study, including drug hypersensitivity findings will be documented in the eCRF as an AE. As a result no summaries or listings will be produced explicitly for physical examinations.

# 11.12 Treatment Compliance

Subjects will be considered to have received a complete dose of IP, and therefore be compliant, if they have received at least 80% of the IP, and cumulative infusion


interruptions (if any) are for no more than a total of 60 minutes. Compliance to IP will be presented for the SAF.

A summary table showing compliance per infusion and overall, by treatment group will be produced.

**Derivation:** Proportion of planned IP is derived from data recorded on the IP eCRF page. Proportion of planned IP will be expressed as a percentage and calculated for each infusion separately as;

Proportion of Planned IP (%) = 
$$\frac{\text{Actual Volume of Infusion (mL)} *}{\text{Planned Volume of Infusion (mL)}} \times 100$$

\* (including resumed dose following interruption for that infusion)

For the purpose of calculation of the proportion of planned IP infused, any missed infusions will be deemed to have an actual volume of infusion set to 0 mL.

Summaries of the timings between infusions (days) by country and overall will also be produced to investigate adherence to the dosing schedule.

## 12 Pharmacokinetic Analyses

# 12.1 Measured and Baseline-Corrected Plasma Apolipoprotein A-I and Phosphatidylcholine Concentrations

Quintiles will produce the following descriptive summaries using the PK Population.

Measured (uncorrected) plasma concentrations and baseline-corrected (change from baseline) concentrations of apoA-I and PC will be listed and summarized by time point, by treatment and by subgroup based on the eGFR (Central) values using central laboratory data.

## 12.2 Population PK Analysis

A population PK analysis using the PK population will be conducted using a separate analysis plan.


## 12.3 Deriving and Summarizing Pharmacokinetic Parameters

A summary of the  $C_{max}$  and the Accumulation Ratios will be produced. These parameters will be calculated as follows:

| Term | Definition |
|---|---|
| Accumulation Ratio $(R_{A)}$ | For subjects receiving CSL112, Accumulation may be obtained using the following accumulation ratio: |
| | $R_A = Baseline\text{-}Corrected \ End \ of \ Infusion_{Infusion \ 1}$ / Baseline-Corrected End of Infusion_{Infusion \ 1} |
| | Note that the Accumulation Ratio will not be calculated for subjects in the Placebo group. |
| Maximum Concentration (C <sub>max</sub> ) | The Maximum Concentration is defined as the End of Infusion concentration after Infusion 1 and Infusion 4. |
| (Cmax) | Both baseline-corrected and measured concentrations will be summarized. |
| | Note that as concentrations are not measured at regular intervals, the end of infusion concentration will serve as the summary for Maximum Concentration. |










### **REFERENCES**

Newcombe, R. Interval estimation for the difference between independent proportions: comparison of eleven methods. Statistics in Medicine, 1998; 17: 873-890.

Price, R., Bonett, D. An improved confidence interval for a linear function of binomial proportions. Computational Statistics & Data Analysis 45, 2004; 449-456.

Guidance for Industry: Drug-Induced Liver Injury: Premarketing Clinical Evaluation. July 2009 http://www.fda.gov/downloads/Drugs/.../Guidances/UCM174090.pdf

Mehran R, Rao SV, Bhatt DL, et al. Standardized bleeding definitions for cardiovascular clinical trials. A consensus report from the Bleeding Academic Research Consortium. Circulation. 2011;123:2736–47.

Stone, NJ et al. 2013 ACC/AHA Guideline on the Treatment of Blood Cholesterol to Reduce Atherosclerotic Cardiovascular Risk in Adults. Journal of the American College of Cardiology 2014; volume 63: No. 25; 2889-2934.


# **Appendices**

# 13.5 List of Tables, Listings, and Figures

## **TABLES**

| Title | Pop. | HL<br>R |
|---|---|---|
| Table 14.1.1.1: Subject Disposition | SCR | HL<br>R |
| Table 14.1.1.2: Enrollment and Randomization by Country and Site | SCR | |
| Table 14.1.1.3: Subject Completion by Visit | SCR | |
| Table 14.1.1.4: Inclusion/Exclusion Criteria | SCR | |
| Table 14.1.1.5: Populations | SCR | |
| Table 14.1.2.1: Major Protocol Deviations | ITT | |
| Table 14.1.2.2: Minor Protocol Deviations | ITT | |
| Table 14.1.3.1: Demographic Characteristics | ITT | HL<br>R |
| Table 14.1.3.2: Subject Baseline Characteristics | ITT | HL<br>R |
| Table 14.1.3.3: Randomization Strata | ITT | |
| Table 14.1.3.4: Agreement of Renal Function by Local and Central Laboratory Assessment | ITT | |
| Table 14.1.3.5.1: Summary of Timings, Overall and by Country | ITT | HL<br>R |
| Table 14.1.3.5.2: Summary of Timings by Type of Index MI | ITT | |
| Table 14.1.3.6: Treatment for Index Myocardial Infarction | ITT | |
| Table 14.1.4.1: Targeted Medical History | ITT | |
| Table 14.1.4.2: Other Medical History, within 3 Months Prior to Screening, by System Organ Class and Preferred Term | ITT | |
| Table 14.1.5: Study Drug Compliance by Infusion | SAF | |
| Table 14.1.6.1: Study Drug Exposure, Overall | SAF | HL<br>R |
| Table 14.1.6.2: Study Drug Exposure, by Infusion | SAF | |
| Table 14.1.6.3: Timings Between Infusions | ITT | |
| Table 14.1.7.1: Prior Medications | ITT | |
| Table 14.1.7.2: Concomitant Medications | ITT | |
| Table 14.1.7.3.1: Medications of Interest Taken the Day Prior to Index MI | ITT | |
| Table 14.1.7.3.2: Medications of Interest Taken the Day Prior to Index MI – Categorical Summary | ITT | |
| Table 14.1.7.4.1: Medications of Interest Taken After Index MI and Continuing at Randomization | ITT | |
| Table 14.1.7.4.2: Medications of Interest Taken After Index MI and Continuing at Randomization – Categorical Summary | ITT | |
| Table 14.1.7.5.1: Medications of Interest Taken as Concomitant Medications | ITT | |
| Table 14.1.7.5.2: Medications of Interest Taken as Concomitant Medications - Categorical Summary | ITT | |
| Table 14.1.7.6: Prior Procedures | ITT | |
| Table 14.1.7.7: Concomitant Procedures | ITT | |
| Table 14.2.1.1: ApoA-I Plasma Concentrations, Measured and Baseline-Corrected Values by Visit and Renal Function | PK | HL<br>R |


| Table 14.2.1.2: Phosphatidylcholine Plasma Concentrations, Measured and Baseline-Corrected Values by Visit, and Renal Function | PK | HL<br>R |
|---|---|---|
| Table 14.2.1.3: Summary of Pharmacokinetic Parameters | PK | HL<br>R |
| CCI | BM | |
| CCI | BM | |
| CCI | BM | |
| CCI | BM | |
| CCI | BM | |
| CCI | BM | |
| CCI | BM | |
| CCI | BM | - |
| CCI | BM | |
| CCI | BM | |
| CCI | BM | |
| Table 14.3.1: Treatment Emergent Adverse Events Overview | SAF | |
| Table 14.3.1.1.1: Treatment Emergent Adverse Events, by System Organ Class and Preferred Term | SAF | |
| Table 14.3.1.1.2: Treatment Emergent Adverse Events, by Preferred Term | SAF | |
| Table 14.3.1.1.3: Treatment Emergent Fatal Adverse Events, by System Organ Class and Preferred Term | SAF | |
| Table 14.3.1.1.4: Treatment Emergent Study Treatment-Related Adverse Events, by System Organ Class and Preferred Term | SAF | |
| Table 14.3.1.1.5: Treatment Emergent Study Treatment-Related Adverse Events, by Preferred Term | SAF | |
| Table 14.3.1.1.6: Treatment-Emergent Study Treatment-Related Fatal AEs by Preferred Term | SAF | |
| Table 14.3.1.1.7: Treatment Emergent Study Procedure-Related Adverse Events, by Preferred Term | SAF | |
| Table 14.3.1.1.8: Treatment Emergent Adverse Events of CTCAE Grade 3 or Higher, by System Organ Class and Preferred Term | SAF | |
| Table 14.3.1.1.9: Treatment Emergent Adverse Events of CTCAE Grade 3 or Higher, by Preferred Term | SAF | |
| Table 14.3.1.1.10: Treatment Emergent Adverse Events Leading to Study Withdrawal, by Preferred Term | SAF | |
| Table 14.3.1.1.11: Treatment Emergent Adverse Events Leading to Permanent Discontinuation of Study Drug, by System Organ Class and Preferred Term | SAF | |
| Table 14.3.1.1.12: Treatment Emergent Adverse Events Leading to Infusion Interruptions, by Preferred Term | SAF | |
| Table 14.3.1.1.13: Treatment Emergent Adverse Events Leading to Infusion Delays, by Preferred Term | SAF | |
| Table 14.3.1.1.14: Treatment Emergent Adverse Events Leading to Skipped Infusions, by Preferred Term | SAF | |
| Table 14.3.1.1.15: Treatment Emergent Adverse Events, by Preferred Term and Maximum Reported CTCAE Grade | SAF | HL<br>R |
| Table 14.3.1.1.16: Treatment Emergent Adverse Events, by Preferred Term and eGFR (Central) Value at the Time of Randomization | SAF | |
| Table 14.3.1.1.17: Treatment Emergent Adverse Events, by Preferred Term and Diabetic Status at the Time of Randomization | SAF | |
| Table 14.3.1.2.1: Treatment Emergent Serious Adverse Events, by System Organ Class and Preferred Term | SAF | HL<br>R |
| Table 14.3.1.2.2: Treatment Emergent Serious Adverse Events, by Preferred Term | SAF | - K |
| Table 14.3.1.2.3: Treatment Emergent Study Treatment-Related Serious Adverse Events, by System Organ Class and Preferred Term | SAF | |
| Table 14.3.1.2.4: Treatment Emergent Study Treatment-Related Serious Adverse Events, by Preferred Term | SAF | |


| Table 14.3.1.3.1: Suspected Adverse Drug Reactions, by System Organ Class and Preferred Term | SAF | HL<br>R |
|---|---|---|
| Table 14.3.1.3.2: Suspected Adverse Drug Reactions, by Preferred Term | SAF | |
| Table 14.3.1.3.3: AESI Overview for Drug Hypersensitivity Reactions | SAF | |
| Table 14.3.1.3.4: Drug Hypersensitivity Reactions, by Preferred Term | SAF | |
| Table 14.3.1.3.5: AESI Overview for Bleeding Events as Reported by Investigators | SAF | |
| Table 14.3.1.3.6: Bleeding Events, as Reported by Investigators, by Preferred Term | SAF | |
| Table 14.3.1.3.7: Summary of Investigator Reported Bleeding Events, by Treatment Group | SAF | HL<br>R |
| Table 14.3.1.3.8: Summary of CEC-Adjudicated Bleeding Events, by Treatment Group | SAF | HL<br>R |
| Table 14.3.1.3.9: AESI Overview for Potential Hemolysis as Identified Using the Haemolytic Disorders SMQ | SAF | |
| Table 14.3.3.1.1: Hematology Assessments (Central Laboratory), Absolute Values and Change from Baseline, by Visit | SAF | HL<br>R |
| Table 14.3.3.1.2: Hematology Assessments (Central Laboratory), Baseline Versus Worst Observation During the Active Treatment Period, Shift Table | SAF | |
| Table 14.3.3.1.3: Summary of Decreases in Hemoglobin ≥ 2 g/dL from Baseline | SAF | HL<br>R |
| Table 14.3.3.2.1: Serum Biochemistry Assessments (Central Laboratory), Absolute Values and Change from Baseline, by Visit | SAF | HL<br>R |
| Table 14.3.3.2.2: Serum Biochemistry Assessments (Central Laboratory), Baseline Versus Worst Observation During the Active Treatment Period, Shift Table | SAF | TC. |
| Table 14.3.3.3.1: Liver Function Assessments (Central Laboratory), Absolute Values and Change from Baseline, by Visit | SAF | HL<br>R |
| Table 14.3.3.3.2: Liver Function Assessments (Central Laboratory), Baseline Versus Worst Observation During the Active Treatment Period, Shift Table | SAF | |
| Table 14.3.3.3.3: Proportion of Subjects with Missing Central Laboratory ALT, Total Bilirubin and Serum Creatinine Results by Visit | SAF | HL<br>R |
| Table 14.3.3.3.4: Summary of Abnormal Liver Function Parameter Values (Sustained for ≥ 24 hours) (Central Laboratory) During the Active Treatment Period | SAF | |
| Table 14.3.3.3.5: Summary of Abnormal Liver Function Parameter Values (Regardless of Confirmation) (Central Laboratory) During the Active Treatment Period | SAF | HL<br>R |
| Table 14.3.3.4.1: Summary of Abnormal Serum Creatinine Values (Central Laboratory) During the Active Treatment Period | SAF | HL<br>R |
| Table 14.3.3.4.2: Summary of Abnormal Serum Creatinine Values (Local Laboratory) During the Active Treatment Period | SAF | HL<br>R |
| Table 14.3.3.5.1: Summary of Urinalysis (Central Laboratory) by Treatment Group and Timepoint | SAF | HL<br>R |
| Table 14.3.3.5.2: Urinalysis (Central Laboratory), Baseline Versus Maximum Observation During the Active Treatment Period, Shift Table | SAF | HL<br>R |
| CCI | SAF | HL<br>R |
| CCI | SAF | |
| CCI | SAF | |
| CCI | SAF | |
| Table 14.3.3.6: Selected CTC Grade 3 and 4 Laboratory Abnormalities (Central Laboratory) | SAF | HL<br>R |
| Table 14.3.3.7: Serum Antibodies to CSL112 and to ApoA-I by Visit | SAF | HL<br>R |
| Table 14.3.4.1.1: Co-Primary Endpoints of Treatment-Emergent Renal SAEs and AKI Events | SAF | HL<br>R |
| Table 14.3.4.1.2: Co-Primary Endpoints of Treatment-Emergent Renal SAEs (CEC-Adjudicated) and AKI Events (Local), Sensitivity Analysis | SAF | HL<br>R |
| Table 14.3.4.1.3: Co-Primary Endpoints of Treatment-Emergent Renal SAEs and AKI Events (Regardless of Confirmation), Sensitivity Analysis | SAF | |
| Table 14.3.4.1.4: Co-Primary Endpoints of Treatment-Emergent Renal SAEs and AKI Events (Excluding Unconfirmed Values), Sensitivity Analysis | SAF | |

## **CSL** Behring

## Statistical Analysis Plan

Protocol Number: CSL112\_2001 Product Name: CSL112

| Table 14.3.4.2.1: Co-Primary Treatment Emergent Investigator Identified Renal SAEs by Preferred Term | SAF | |
|---|---|---|
| Table 14.3.4.2.2: Co-Primary Treatment Emergent CEC-Adjudicated Renal SAEs by Preferred Term | SAF | |
| Table 14.3.4.2.3: Co-Primary Positively Adjudicated Treatment Related Renal SAEs by Preferred Term | SAF | |
| Table 14.3.4.2.4: Co-Primary Treatment Emergent Renal SAEs (CEC-Adjudicated), by Preferred Term and Adjudication Details | SAF | |
| Table 14.3.4.2.5: Co-Primary Exploratory Summary of the Renal Safety Endpoint, by Subgroup | SAF | HL<br>R |
| Table 14.3.4.2.6: Summary of CEC-Adjudicated Serious Renal Events, by Treatment Group | SAF | HL<br>R |
| Table 14.3.4.3.1: Co-Primary Summary of Treatment-Emergent AKI events | SAF | HL<br>R |
| Table 14.3.4.3.2: Comparison of AKI Rates Based on the Timing of Serum Creatinine Determinations for Dosing Eligibility | SAF | HL<br>R |
| Table 14.3.5.1: Vital Signs Variables, Absolute Values and Change from Baseline, by Visit | SAF | |
| Table 14.3.5.2: Incidence of Treatment-Emergent Markedly Abnormal Vital Signs, Treatment-Emergent Changes | SAF | |
| Table 14.3.6.1: ECG Variables, Absolute Values and Change from Baseline, by Visit | SAF | |
| Table 14.3.6.2: ECG, Baseline Versus Last Assessment During the Active Treatment Period, Shift Table | SAF | |
| Table 14.3.6.3: Incidence of Treatment-Emergent Markedly Abnormal ECG Intervals | SAF | |
| Table 14.3.6.4: Overall Interpretation of ECG Results by Visit | SAF | |


#### **FIGURES**

| Title | Pop. | HLR |
|---|---|---|
| Figure 14.3.3.2.3.1: Box Plots of eGFR (Central) Values by Visit and Treatment | SAF | |
| Figure 14.3.3.2.3.2: Box Plots of eGFR (Central) Values by Visit, Treatment and Renal Function | SAF | |
| Figure 14.3.3.2.4: Box Plots of eGFR (Central) Change from Baseline by Visit and Treatment | SAF | |
| Figure 14.3.3.2.5: Box Plots of eGFR (Central) Change from Baseline by Visit, Treatment and Renal Function | SAF | |
| CCI | SAF | |
| Figure 14.3.3.4.3.1: Box Plots of ALT Values (Central Laboratory) by Visit and Treatment | SAF | |
| Figure 14.3.3.4.3.2: Box Plots of ALT xULN Values (Central Laboratory) by Visit and Treatment | SAF | |
| Figure 14.3.3.4.4.1: Box Plots of Total Bilirubin Values (Central Laboratory) by Visit and Treatment | SAF | |
| Figure 14.3.3.4.4.2: Box Plots of Total Bilirubin xULN Values (Central Laboratory) by Visit and Treatment | SAF | |
| Figure 14.3.3.4.5: Box Plots of Direct Bilirubin xULN Values (Central Laboratory) by Visit and Treatment | SAF | |
| Figure 14.3.3.4.6.1: Box Plots of Serum Creatinine Values (Central Laboratory) by Visit and Treatment | SAF | |
| Figure 14.3.3.4.6.2: Box Plots of Serum Creatinine Values (Central Laboratory) by Visit, Treatment and Renal Function | SAF | |
| Figure 14.3.3.4.6.3: Box Plots of Serum Creatinine Change from Baseline Values (Central Laboratory) by Visit and Treatment | SAF | |
| Figure 14.3.3.4.7: Plot of Total Bilirubin vs ALT xULN Values (Central Laboratory) by Treatment – All Subjects | SAF | |
| Figure 14.3.3.4.8: Plot of Total Bilirubin vs ALT xULN Values (Central Laboratory) by Treatment – Excluding Subjects with a History of Gilberts Syndrome | SAF | |
| Figure 14.3.3.4.9: Plot of Total Bilirubin vs AST xULN Values (Central Laboratory) by Treatment – All Subjects | SAF | |
| Figure 14.3.3.4.10: Plot of Total Bilirubin vs AST xULN Values (Central Laboratory) by Treatment – Excluding Subjects with a History of Gilberts Syndrome | SAF | |
| Figure 14.3.3.4.11: Individual Series Plots of Serum Creatinine Over Time for Subjects with Any Central Laboratory Change from Baseline $\geq 0.3 \text{mg/dL}$ | SAF | |
| Figure 14.3.5.3: Box Plots of Systolic Blood Pressure Change from Baseline by Visit and Treatment | SAF | |
| Figure 14.3.5.4: Box Plots of Diastolic Blood Pressure Change from Baseline by Visit and Treatment | SAF | |
| Figure 14.3.5.5: Box Plots of Pulse Change from Baseline by Visit and Treatment | SAF | |


#### LISTINGS

| Title | Pop. | HLR |
|---|---|---|
| Listing 14.3.2.1: Fatal Adverse Events | SAF | |
| Listing 14.3.2.2: Deaths Among Subjects Who were Screened but Not Treated | SCR | |
| Listing 16.2.1.1: Subject Disposition | ITT | |
| Listing 16.2.1.2: Subject Completion by Visit | SCR | |
| Listing 16.2.1.3: Other Disposition | ITT | |
| Listing 16.2.1.4: Screen Failures | SCR | |
| Listing 16.2.1.5 Final Subject Status | ITT | |
| Listing 16.2.1.6: Enrollment of Treated Subjects by Country and by Site | SAF | |
| Listing 16.2.2.1: Protocol Deviations | ITT | |
| Listing 16.2.2.2: Protocol Deviations Related to Infusion Duration | SAF | |
| Listing 16.2.2.3: Eligibility Criteria Compliance | SCR | |
| Listing 16.2.2.4: Randomized and Actual Treatments | ITT | |
| Listing 16.2.2.5: Difference Between the Strata Allocation based on eGFR within the IRT System vs eGFR Derived from Central Laboratory | ITT | |
| Listing 16.2.2.6: Incorrect Strata Allocation based on eGFR within the IRT System vs eGFR Derived from Local Laboratory | ITT | |
| Listing 16.2.2.7: Incorrect Strata Allocation based on Medical History of Diabetes within the IRT System vs Data Reported on eCRF | ITT | |
| Listing 16.2.2.8: Timings | ITT | |
| Listing 16.2.3.1: Analysis Populations | SCR | |
| | SAF | |
| Listing 16.2.4.1: Demographic Characteristics | ITT | |
| Listing 16.2.4.2.1: Other Baseline Characteristics - Index Myocardial Infarction | ITT | |
| Listing 16.2.4.2.2: Other Baseline Characteristics - Pregnancy Test Results | ITT | |
| Listing 16.2.4.2.3: Other Baseline Characteristics - FSH Measurements | ITT | |
| Listing 16.2.4.3.1: Targeted Medical History | ITT | |
| Listing 16.2.4.3.2: Other Medical History | ITT | |
| Listing 16.2.4.4.1: Prior Medication | ITT | |
| Listing 16.2.4.4.2: Concomitant Medications | ITT | |
| Listing 16.2.4.4.3: Medications of Interest Taken Prior to Index MI | ITT | |
| Listing 16.2.4.4.4: Medications of Interest Taken After Index MI and Continuing at Randomization | ITT | |
| Listing 16.2.4.4.5: Medications of Interest Taken as Concomitant Medications | ITT | |
| Listing 16.2.4.4.6: Concomitant or Prior Procedures | ITT | |
| Listing 16.2.4.4.7: Post Treatment Procedures | ITT | |
| Listing 16.2.4.4.8: Use of Renal Replacement Therapy | ITT | |
| Listing 16.2.5.1: Study Drug Exposure and Compliance | SAF | |
| Listing 16.2.5.2: Infusion Interruptions | SAF | |
| Listing 16.2.5.3: Overdoses | SAF | |


| Listing 16.2.6.1: Plasma Concentrations to ApoA-I and PC | PK |
|---|---|
| Listing 16.2.6.2: Pharmacokinetic Parameters | PK |
| CCI | BM |
| CCI | BM |
| CCI | BM |
| CCI | BM |
| Listing 16.2.7.1.1: Adverse Events | SAF |
| Listing 16.2.7.1.2: Adverse Events, by Treatment Group and Subjects Experiencing the Preferred Terms | SAF |
| Listing 16.2.7.1.3: Adverse Events of CTCAE Grade 3 or Higher | SAF |
| Listing 16.2.7.1.4: Adverse Events Leading to Withdrawal from the Study | SAF |
| Listing 16.2.7.1.5: Adverse Events Leading to Permanent Discontinuation of Study Treatment | SAF |
| Listing 16.2.7.1.6: Adverse Events Leading to Infusion Interruptions | SAF |
| Listing 16.2.7.1.7: Adverse Events Leading to Infusion Delays | SAF |
| Listing 16.2.7.1.8: Adverse Events Leading to Skipped Infusions | SAF |
| Listing 16.2.7.1.9: Adverse Events as Identified by Investigators on the Serious Renal Event CRF Page | SCR |
| Listing 16.2.7.1.10: Adverse Events Among Subjects Who were Screened but Not Treated | SCR |
| Listing 16.2.7.2: Serious Adverse Events | SAF |
| Listing 16.2.7.3.1: Adverse Drug Reactions | SAF |
| Listing 16.2.7.3.2: AESI - Drug Hypersensitivity Reactions | SAF |
| Listing 16.2.7.3.3: AESI - Hemolysis as Identifed Using the Haemolytic Disorders SMQ | SAF |
| Listing 16.2.7.3.4.1: AESI – Bleeding Events | SAF |
| Listing 16.2.7.3.4.2: Endpoint Bleeding Events as Reported by Investigators | SAF |
| Listing 16.2.7.3.4.3: Endpoint Bleeding Events (CEC-Adjudicated) | SAF |
| Listing 16.2.7.4.1: Endpoint Serious Renal Events as Reported by Investigators | SAF |
| Listing 16.2.7.4.2: Endpoint Serious Renal Events (CEC-Adjudicated) | SAF |
| Listing 16.2.8.1.1.1: Hematology (Central Laboratory) | SAF |
| Listing 16.2.8.1.1.2: Hematology (Local Laboratory) | SAF |
| Listing 16.2.8.1.2.1: Central Laboratory Values Outside Normal Reference Ranges - Hematology | SAF |
| Listing 16.2.8.1.2.2: Local Laboratory Values Outside Normal Reference Ranges - Hematology | SAF |
| Listing 16.2.8.1.3.1: CTC Grade 3 and 4 Laboratory Abnormalities (Central Laboratory) - Hematology | SAF |
| Listing 16.2.8.1.3.2: CTC Grade 3 and 4 Laboratory Abnormalities (Local Laboratory) - Hematology | SAF |
| Listing 16.2.8.1.4: Hematology Assessments for Subjects with Potential Hemolysis Identified by Decreases in Hemoglobin $\geq$ 2 g/dL from Baseline | SAF |
| Listing 16.2.8.1.5: Investigations Following Potential Hemolysis as Identified by Investigators | SAF |
| Listing 16.2.8.2.1.1: Serum Biochemistry (Central Laboratory) | SAF |
| Listing 16.2.8.2.1.2: Serum Biochemistry (Local Laboratory) | SAF |
| Listing 16.2.8.2.2.1: Central Laboratory Values Outside Normal Reference Ranges - Serum Biochemistry | SAF |
| Listing 16.2.8.2.2.2: Local Laboratory Values Outside Normal Reference Ranges - Serum Biochemistry | SAF |
| Listing 16.2.8.2.3.1: CTC Grade 3 and 4 Laboratory Abnormalities (Central Laboratory) - Serum Biochemistry | SAF |


## **CSL** Behring

## Statistical Analysis Plan

Protocol Number: CSL112\_2001 Product Name: CSL112

| Listing 16.2.8.2.4: Co-Primary AKI Events Listing 16.2.8.2.5: Serum Creatinine (Central Laboratory) for Subjects with either Treatment-Emergent Renal SAEs or AKI SAF HLR Listing 16.2.8.2.6: Serum Creatinine (Central Laboratory) for Subjects with either Treatment-Emergent Renal SAEs or AKI SAF HLR Events (Regardless of Confirmation) Listing 16.2.8.3.1.1: Liver Function (Central Laboratory) SAF Listing 16.2.8.3.1.2: Liver Function (Local Laboratory) SAF Listing 16.2.8.3.1.2: Liver Function (Local Laboratory) Listing 16.2.8.3.2: Liver Function (Local Laboratory) Listing 16.2.8.3.3.1: CTC Grade 3 and 4 Laboratory Abnormal Reference Ranges - Liver Function SAF Listing 16.2.8.3.3.2: CTC Grade 3 and 4 Laboratory Abnormalities (Central Laboratory) - Liver Function SAF Listing 16.2.8.3.3.1: Liver Function Parameters (Central Laboratory) - Liver Function SAF Listing 16.2.8.3.4.1: Liver Function Parameters (Central Laboratory) for Subjects with Any Abnormal Liver Function SAF Listing 16.2.8.3.4.2: Liver Function Parameters (Local Laboratory) for Subjects with Any Abnormal Liver Function SAF Listing 16.2.8.3.5.1: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Sacinatory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) SAF Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) SAF Listing 16.2.8.3.9: Local Laboratory Serum Creatinine Values (µmol/L) Pre and Post-Contrast Agent SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.4.1: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.1: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.1: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.1: Urinalysis Additional Testing SAF Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.9.1: Vital Signs Treatment-Emergent V | | | |
|---|---|---|---|
| Listing 16.2.8.2.5: Serum Creatinine (Central Laboratory) for Subjects with either Treatment-Emergent Renal SAEs or AKI Events (Regardless of Confirmation) Listing 16.2.8.2.6: Serum Creatinine (Central Laboratory) for Subjects with either Treatment-Emergent Renal SAEs or AKI Events (Regardless of Confirmation) SAF Listing 16.2.8.3.1.1: Liver Function (Central Laboratory) SAF Listing 16.2.8.3.1.2: Liver Function (Local Laboratory) Listing 16.2.8.3.1.2: Liver Function (Local Laboratory) Listing 16.2.8.3.1.2: Liver Function (Local Laboratory) Listing 16.2.8.3.1.2: Liver Function (Local Laboratory) Listing 16.2.8.3.3.1: CTC Grade 3 and 4 Laboratory Abnormal Reference Ranges - Liver Function SAF Listing 16.2.8.3.3.1: CTC Grade 3 and 4 Laboratory Abnormalities (Central Laboratory) - Liver Function SAF Listing 16.2.8.3.3.1: Liver Function Parameters (Central Laboratory) for Subjects with Any Abnormal Liver Function SAF Assessments Listing 16.2.8.3.4.1: Liver Function Parameters (Central Laboratory) for Subjects with Any Abnormal Liver Function SAF Assessments Listing 16.2.8.3.5.1: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Central Laboratory) Critera Met Listing 16.2.8.3.5.2: Local Laboratory Serum Creatinine Values (µmol/L) Pre and Post-Contrast Agent SAF Listing 16.2.8.3.5: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.4.1: Urinalysis (Central Laboratory) Listing 16.2.8.4.1: Urinalysis (Local Laboratory) Listing 16.2.8.4.1: Urinalysis Additional Testing Listing 16.2.8.3: Hepatic Injury Assessments SAF Listing 16.2.8.3: Hepatic Injury Assessments Listing 16.2.8.1: Vital Signs Listing 16.2.9: | Listing 16.2.8.2.3.2: CTC Grade 3 and 4 Laboratory Abnormalities (Local Laboratory) - Serum Biochemistry | SAF | |
| Events Events Events (Regardless of Confirmation) Listing 16.2.8.2.6: Serum Creatinine (Central Laboratory) for Subjects with either Treatment-Emergent Renal SAEs or AKI Events (Regardless of Confirmation) Listing 16.2.8.3.1.1: Livier Function (Local Laboratory) SAF Listing 16.2.8.3.1.2: Livier Function (Local Laboratory) SAF Listing 16.2.8.3.2.1: Central Laboratory Values Outside Normal Reference Ranges - Liver Function SAF Listing 16.2.8.3.3.1: CTC Grade 3 and 4 Laboratory Abnormal Reference Ranges - Liver Function SAF Listing 16.2.8.3.3.1: CTC Grade 3 and 4 Laboratory Abnormalities (Central Laboratory) - Liver Function SAF Listing 16.2.8.3.4.1: Liver Function Parameters (Central Laboratory) for Subjects with Any Abnormal Liver Function SAF SAF Listing 16.2.8.3.4.1: Liver Function Parameters (Cocal Laboratory) for Subjects with Any Abnormal Liver Function SAF SAF Listing 16.2.8.3.5.1: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) Central Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.5.1: Serum Creatinine Central Laboratory) Critera Met Listing 16.2.8.3.5.1: Cocal Laboratory Serum Creatinine Values (μmol/L) Pre and Post-Contrast Agent SAF Listing 16.2.8.3.5.1: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.3.5: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.4.1.1: Urinalysis (Central Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis Additional Testing SAF Listing 16.2.8.4.1.1: Urinalysis Additional Testing Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.9.1: Vital Signs Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF | Listing 16.2.8.2.4: Co-Primary AKI Events | SAF | |
| Events (Regardless of Confirmation) Listing 16.2.8.3.1.1: Liver Function (Central Laboratory) SAF Listing 16.2.8.3.1.2: Liver Function (Local Laboratory) SAF Listing 16.2.8.3.2.1: Central Laboratory Values Outside Normal Reference Ranges - Liver Function SAF Listing 16.2.8.3.2.2: Local Laboratory Values Outside Normal Reference Ranges - Liver Function SAF Listing 16.2.8.3.3.1: CTC Grade 3 and 4 Laboratory Abnormalities (Central Laboratory) - Liver Function SAF Listing 16.2.8.3.3.1: CTC Grade 3 and 4 Laboratory Abnormalities (Local Laboratory) - Liver Function SAF Listing 16.2.8.3.4.1: Liver Function Parameters (Central Laboratory) for Subjects with Any Abnormal Liver Function SAF Listing 16.2.8.3.4.2: Liver Function Parameters (Local Laboratory) for Subjects with Any Abnormal Liver Function SAF Assessments Listing 16.2.8.3.4.2: Liver Function Parameters (Local Laboratory) for Subjects with Any Abnormal Liver Function SAF Assessments Listing 16.2.8.3.5.1: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) Central Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.5.1: Local Laboratory Serum Creatinine Values (µmol/L) Pre and Post-Contrast Agent SAF Listing 16.2.8.3.5: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.4.1.1: Urinalysis (Central Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis Additional Testing Listing 16.2.8.5: Hepatic Injury Assessments Listing 16.2.8.6: Investigations Following Drug Hypersensitivity Listing 16.2.8.6: Investigations Following Drug Hypersensitivity Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-1 Listing 16.2.9.1: Vital Signs Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF | Listing 16.2.8.2.5: Serum Creatinine (Central Laboratory) for Subjects with either Treatment-Emergent Renal SAEs or AKI Events | SAF | HLR |
| Listing 16.2.8.3.1.2: Liver Function (Local Laboratory) Listing 16.2.8.3.2.1: Central Laboratory Values Outside Normal Reference Ranges - Liver Function SAF Listing 16.2.8.3.2.2: Local Laboratory Values Outside Normal Reference Ranges - Liver Function SAF Listing 16.2.8.3.3.1: CTC Grade 3 and 4 Laboratory Abnormalities (Central Laboratory) - Liver Function SAF Listing 16.2.8.3.3.2: CTC Grade 3 and 4 Laboratory Abnormalities (Local Laboratory) - Liver Function SAF Listing 16.2.8.3.3.1: Liver Function Parameters (Central Laboratory) for Subjects with Any Abnormal Liver Function SAF Listing 16.2.8.3.4.2: Liver Function Parameters (Local Laboratory) for Subjects with Any Abnormal Liver Function SAF Listing 16.2.8.3.4.2: Liver Function Parameters (Local Laboratory) for Subjects with Any Abnormal Liver Function SAF Listing 16.2.8.3.5.1: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) Central Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.5: Summary of Serum Creatinine (Central Laboratory) Critera Met Listing 16.2.8.3.7: Local Laboratory Serum Creatinine Values (μmol/L) Pre and Post-Contrast Agent SAF Listing 16.2.8.3.8: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.4.1.1: Urinalysis (Central Laboratory) SAF Listing 16.2.8.4.2: Urinalysis Additional Testing SAF Listing 16.2.8.4.2: Urinalysis Additional Testing SAF Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-1 SAF Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF | Listing 16.2.8.2.6: Serum Creatinine (Central Laboratory) for Subjects with either Treatment-Emergent Renal SAEs or AKI Events (Regardless of Confirmation) | SAF | HLR |
| Listing 16.2.8.3.2.1: Central Laboratory Values Outside Normal Reference Ranges - Liver Function SAF Listing 16.2.8.3.2.2: Local Laboratory Values Outside Normal Reference Ranges - Liver Function SAF Listing 16.2.8.3.3.1: CTC Grade 3 and 4 Laboratory Abnormalities (Central Laboratory) - Liver Function SAF Listing 16.2.8.3.3.2: CTC Grade 3 and 4 Laboratory Abnormalities (Local Laboratory) - Liver Function SAF Listing 16.2.8.3.4.1: Liver Function Parameters (Central Laboratory) for Subjects with Any Abnormal Liver Function SAF Listing 16.2.8.3.4.2: Liver Function Parameters (Local Laboratory) for Subjects with Any Abnormal Liver Function SAF Listing 16.2.8.3.5.1: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) Central Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.5: Summary of Serum Creatinine (Central Laboratory) Critera Met Listing 16.2.8.3.7: Local Laboratory Serum Creatinine Values (µmol/L) Pre and Post-Contrast Agent SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.4.1.1: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis Additional Testing SAF Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-1 SAF Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.1: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.1.1: 12-Lead ECG SAF | Listing 16.2.8.3.1.1: Liver Function (Central Laboratory) | SAF | |
| Listing 16.2.8.3.2.2: Local Laboratory Values Outside Normal Reference Ranges - Liver Function SAF Listing 16.2.8.3.3.1: CTC Grade 3 and 4 Laboratory Abnormalities (Central Laboratory) - Liver Function SAF Listing 16.2.8.3.4.1: Liver Function Parameters (Central Laboratory) for Subjects with Any Abnormal Liver Function SAF Listing 16.2.8.3.4.1: Liver Function Parameters (Central Laboratory) for Subjects with Any Abnormal Liver Function SAF Assessments Listing 16.2.8.3.4.2: Liver Function Parameters (Local Laboratory) for Subjects with Any Abnormal Liver Function SAF Listing 16.2.8.3.5.1: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Central Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine (Central Laboratory) Critera Met Listing 16.2.8.3.6: Summary of Serum Creatinine Values (µmol/L) Pre and Post-Contrast Agent SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.4.1.1: Urinalysis (Central Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis Additional Testing SAF Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.1.1: 12-Lead ECG | Listing 16.2.8.3.1.2: Liver Function (Local Laboratory) | SAF | |
| Listing 16.2.8.3.3.1: CTC Grade 3 and 4 Laboratory Abnormalities (Central Laboratory) - Liver Function SAF Listing 16.2.8.3.4.1: Liver Function Parameters (Central Laboratory) of Subjects with Any Abnormal Liver Function SAF Listing 16.2.8.3.4.1: Liver Function Parameters (Central Laboratory) for Subjects with Any Abnormal Liver Function SAF Assessments Listing 16.2.8.3.4.2: Liver Function Parameters (Local Laboratory) for Subjects with Any Abnormal Liver Function SAF Assessments Listing 16.2.8.3.4.2: Liver Function Parameters (Local Laboratory) for Subjects with Any Abnormal Liver Function SAF Listing 16.2.8.3.5.1: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Central Laboratory) Critera Met Listing 16.2.8.3.6: Summary of Serum Creatinine (Central Laboratory) Critera Met Listing 16.2.8.3.7: Local Laboratory Serum Creatinine Values (μmol/L) Pre and Post-Contrast Agent SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.4.1.1: Urinalysis (Central Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-1 SAF Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.1.1: 12-Lead ECG SAF | Listing 16.2.8.3.2.1: Central Laboratory Values Outside Normal Reference Ranges - Liver Function | SAF | |
| Listing 16.2.8.3.3.2: CTC Grade 3 and 4 Laboratory Abnormalities (Local Laboratory) - Liver Function SAF Listing 16.2.8.3.4.1: Liver Function Parameters (Central Laboratory) for Subjects with Any Abnormal Liver Function Assessments Listing 16.2.8.3.4.2: Liver Function Parameters (Local Laboratory) for Subjects with Any Abnormal Liver Function SAF Assessments Listing 16.2.8.3.5.1: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Central Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Central Laboratory) Critera Met SAF Listing 16.2.8.3.7: Local Laboratory Serum Creatinine Values (µmol/L) Pre and Post-Contrast Agent SAF Listing 16.2.8.3.8: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.4.1.1: Urinalysis (Central Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) SAF Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-I Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.10.1: 12-Lead ECG SAF | Listing 16.2.8.3.2.2: Local Laboratory Values Outside Normal Reference Ranges - Liver Function | SAF | |
| Listing 16.2.8.3.4.1: Liver Function Parameters (Central Laboratory) for Subjects with Any Abnormal Liver Function Assessments SAF Listing 16.2.8.3.4.2: Liver Function Parameters (Local Laboratory) for Subjects with Any Abnormal Liver Function Assessments Listing 16.2.8.3.5.1: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Central Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.5: Local Laboratory Serum Creatinine (Central Laboratory) Critera Met SAF Listing 16.2.8.3.7: Local Laboratory Serum Creatinine Values (μποl/L) Pre and Post-Contrast Agent SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory eGFR Values SAF Listing 16.2.8.4.1.1: Urinalysis (Central Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) SAF Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-I Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.10.1: 12-Lead ECG SAF | Listing 16.2.8.3.3.1: CTC Grade 3 and 4 Laboratory Abnormalities (Central Laboratory) - Liver Function | SAF | |
| Assessments Listing 16.2.8.3.4.2: Liver Function Parameters (Local Laboratory) for Subjects with Any Abnormal Liver Function Assessments Listing 16.2.8.3.5.1: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Central Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.6: Summary of Serum Creatinine (Central Laboratory) Critera Met Listing 16.2.8.3.7: Local Laboratory Serum Creatinine Values (μmol/L) Pre and Post-Contrast Agent SAF Listing 16.2.8.3.8: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory eGFR Values SAF Listing 16.2.8.4.1.1: Urinalysis (Central Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.2: Urinalysis Additional Testing SAF Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-I SAF Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.10.1: 12-Lead ECG SAF | Listing 16.2.8.3.3.2: CTC Grade 3 and 4 Laboratory Abnormalities (Local Laboratory) - Liver Function | SAF | |
| Assessments Listing 16.2.8.3.5.1: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) C(central Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.6: Summary of Serum Creatinine (Central Laboratory) Critera Met SAF Listing 16.2.8.3.7: Local Laboratory Serum Creatinine Values (µmol/L) Pre and Post-Contrast Agent SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory eGFR Values SAF Listing 16.2.8.4.1.1: Urinalysis (Central Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis Additional Testing SAF Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-I SAF Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.9.1: 12-Lead ECG SAF | Listing 16.2.8.3.4.1: Liver Function Parameters (Central Laboratory) for Subjects with Any Abnormal Liver Function Assessments | SAF | |
| (Central Laboratory) Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI (≥ 3x Baseline or ≥ 4.0mg/dL) (Local Laboratory) Listing 16.2.8.3.6: Summary of Serum Creatinine (Central Laboratory) Critera Met SAF Listing 16.2.8.3.7: Local Laboratory Serum Creatinine Values (μmol/L) Pre and Post-Contrast Agent SAF Listing 16.2.8.3.8: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory eGFR Values SAF Listing 16.2.8.4.1.1: Urinalysis (Central Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.2: Urinalysis Additional Testing SAF Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-I SAF Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF | Listing 16.2.8.3.4.2: Liver Function Parameters (Local Laboratory) for Subjects with Any Abnormal Liver Function Assessments | SAF | |
| Laboratory) Listing 16.2.8.3.6: Summary of Serum Creatinine (Central Laboratory) Critera Met Listing 16.2.8.3.7: Local Laboratory Serum Creatinine Values (μmol/L) Pre and Post-Contrast Agent Listing 16.2.8.3.8: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory eGFR Values SAF Listing 16.2.8.4.1.1: Urinalysis (Central Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.2: Urinalysis Additional Testing SAF Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-I Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.10.1: 12-Lead ECG | Listing 16.2.8.3.5.1: Serum Creatinine Assessments for Subjects with a Stage 3 AKI ( $\ge 3x$ Baseline or $\ge 4.0$ mg/dL) (Central Laboratory) | SAF | |
| Listing 16.2.8.3.7: Local Laboratory Serum Creatinine Values (µmol/L) Pre and Post-Contrast Agent Listing 16.2.8.3.8: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory eGFR Values SAF Listing 16.2.8.4.1.1: Urinalysis (Central Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.2: Urinalysis Additional Testing SAF Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-I SAF Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.10.1: 12-Lead ECG | Listing 16.2.8.3.5.2: Serum Creatinine Assessments for Subjects with a Stage 3 AKI ( $\ge 3x$ Baseline or $\ge 4.0$ mg/dL) (Local Laboratory) | SAF | |
| Listing 16.2.8.3.8: Local Laboratory vs. Central Laboratory Serum Creatinine Samples SAF Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory eGFR Values SAF Listing 16.2.8.4.1.1: Urinalysis (Central Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.2: Urinalysis Additional Testing SAF Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-I Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.10.1: 12-Lead ECG SAF | Listing 16.2.8.3.6: Summary of Serum Creatinine (Central Laboratory) Critera Met | SAF | |
| Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory eGFR Values Listing 16.2.8.4.1.1: Urinalysis (Central Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.2: Urinalysis Additional Testing SAF Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-I Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.10.1: 12-Lead ECG SAF | Listing 16.2.8.3.7: Local Laboratory Serum Creatinine Values (µmol/L) Pre and Post-Contrast Agent | SAF | |
| Listing 16.2.8.4.1.1: Urinalysis (Central Laboratory) SAF Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.2: Urinalysis Additional Testing SAF Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-I SAF Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.10.1: 12-Lead ECG SAF | Listing 16.2.8.3.8: Local Laboratory vs. Central Laboratory Serum Creatinine Samples | SAF | HLR |
| Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) SAF Listing 16.2.8.4.2: Urinalysis Additional Testing SAF Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-I Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.10.1: 12-Lead ECG SAF | Listing 16.2.8.3.9: Local Laboratory vs. Central Laboratory eGFR Values | SAF | |
| Listing 16.2.8.4.2: Urinalysis Additional Testing SAF Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-I Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.10.1: 12-Lead ECG SAF | Listing 16.2.8.4.1.1: Urinalysis (Central Laboratory) | SAF | |
| Listing 16.2.8.5: Hepatic Injury Assessments SAF Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-I Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.10.1: 12-Lead ECG SAF | Listing 16.2.8.4.1.2: Urinalysis (Local Laboratory) | SAF | |
| Listing 16.2.8.6: Investigations Following Drug Hypersensitivity SAF Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-I Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.10.1: 12-Lead ECG SAF | Listing 16.2.8.4.2: Urinalysis Additional Testing | SAF | |
| Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-I Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.10.1: 12-Lead ECG SAF | Listing 16.2.8.5: Hepatic Injury Assessments | SAF | |
| Listing 16.2.9.1: Vital Signs SAF Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.10.1: 12-Lead ECG SAF | Listing 16.2.8.6: Investigations Following Drug Hypersensitivity | SAF | |
| Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria SAF Listing 16.2.10.1: 12-Lead ECG SAF | Listing 16.2.8.7: Serum Antibody Reciprocal Titer to CSL112 and to ApoA-I | SAF | |
| Listing 16.2.10.1: 12-Lead ECG SAF | Listing 16.2.9.1: Vital Signs | SAF | |
| | Listing 16.2.9.2: Vital Signs, Treatment-Emergent Values Meeting Markedly Abnormal Criteria | SAF | |
| Listing 16.2.10.2: Abnormal ECG - Overall Evaluation SAF | Listing 16.2.10.1: 12-Lead ECG | SAF | |
| 215th g 10/2110/21110101that 200 0 10th 2 throat 200 | Listing 16.2.10.2: Abnormal ECG - Overall Evaluation | SAF | |


## 13.6 List of Preferred Terms within Standardised MedDRA Queries

## 13.6.1 Co-Primary Endpoint Renal SAEs

| MedDRA v20.0 SMQ | SMQ<br>Code | PT | PT Code |
|---|---|---|---|
| Acute Renal Failure, Narrow | 20000003 | Acute kidney injury | 10069339 |
| | | Acute phosphate nephropathy | 10069688 |
| | | Acute prerenal failure | 10001017 |
| | | Anuria | 10002847 |
| | | Azotaemia | 10003885 |
| | | Continuous haemodiafiltration | 10066338 |
| | | Dialysis | 10061105 |
| | | Foetal renal impairment | 10078987 |
| | | Haemodialysis | 10018875 |
| | | Haemofiltration | 10053090 |
| | | Hyponatriuria | 10077515 |
| | | Neonatal anuria | 10049778 |
| | | Nephropathy toxic | 10029155 |
| | | Oliguria | 10030302 |
| | | Peritoneal dialysis | 10034660 |
| | | Prerenal failure | 10072370 |
| | | Renal failure | 10038435 |
| | | Renal failure neonatal | 10038447 |
| | | Renal impairment | 10062237 |
| | | Renal impairment neonatal | 10049776 |


# 13.6.2 Drug Hypersensitivity

| MedDRA v20.0 SMQ | SMQ Code | PT | PT Code |
|---|---|---|---|
| Hypersensitivity, Narrow | 20000214 | Acute generalised exanthematous pustulosis | 10048799 |
| | | Administration site dermatitis | 10075096 |
| | | Administration site eczema | 10075099 |
| | | Administration site hypersensitivity | 10075102 |
| | | Administration site rash | 10071156 |
| | | Administration site recall reaction | 10075964 |
| | | Administration site urticaria | 10075109 |
| | | Administration site vasculitis | 10075969 |
| | | Allergic bronchitis | 10052613 |
| | | Allergic colitis | 10059447 |
| | | Allergic cough | 10053779 |
| | | Allergic cystitis | 10051394 |
| | | Allergic eosinophilia | 10075185 |
| | | Allergic gastroenteritis | 10075308 |
| | | Allergic hepatitis | 10071198 |
| | | Allergic keratitis | 10057380 |
| | | Allergic myocarditis | 10001715 |
| | | Allergic oedema | 10060934 |
| | | Allergic otitis externa | 10075072 |
| | | Allergic otitis media | 10061557 |
| | | Allergic pharyngitis | 10050639 |
| | | Allergic reaction to excipient | 10078853 |
| | | Allergic respiratory disease | 10063532 |
| | | Allergic respiratory symptom | 10063527 |
| | | Allergic sinusitis | 10049153 |
| | | Allergic transfusion reaction | 10066173 |
| | | Allergy alert test positive | 10075479 |
| | | Allergy test positive | 10056352 |
| | | Allergy to immunoglobulin therapy | 10074079 |
| | | Allergy to surgical sutures | 10077279 |
| | | Allergy to vaccine | 10055048 |
| | | Alveolitis allergic | 10001890 |
| | | Anaphylactic reaction | 10002198 |
| | | Anaphylactic shock | 10002199 |


| Anaphylactic transfusion reaction | 10067113 |
|-----------------------------------------------|----------|
| Anaphylactoid reaction | 10002216 |
| Anaphylactoid shock | 10063119 |
| Anaphylaxis treatment | 10002222 |
| Angioedema | 10002424 |
| Antiallergic therapy | 10064059 |
| Antiendomysial antibody positive | 10065514 |
| Anti-neutrophil cytoplasmic antibody positive | 10050894 |
| vasculitis | |
| Application site dermatitis | 10003036 |
| Application site eczema | 10050099 |
| Application site hypersensitivity | 10063683 |
| Application site rash | 10003054 |
| Application site recall reaction | 10076024 |
| Application site urticaria | 10050104 |
| Application site vasculitis | 10076027 |
| Arthritis allergic | 10061430 |
| Aspirin-exacerbated respiratory disease | 10075084 |
| Atopy | 10003645 |
| Blepharitis allergic | 10005149 |
| Blood immunoglobulin E abnormal | 10005589 |
| Blood immunoglobulin E increased | 10005591 |
| Bromoderma | 10006404 |
| Bronchospasm | 10006482 |
| Catheter site dermatitis | 10073992 |
| Catheter site eczema | 10073995 |
| Catheter site hypersensitivity | 10073998 |
| Catheter site rash | 10052271 |
| Catheter site urticaria | 10052272 |
| Catheter site vasculitis | 10074014 |
| Chronic eosinophilic rhinosinusitis | 10071399 |
| Chronic hyperplastic eosinophilic sinusitis | 10071380 |
| Circulatory collapse | 10009192 |
| Circumoral oedema | 10052250 |
| Conjunctival oedema | 10010726 |
| Conjunctivitis allergic | 10010744 |


| <br> | |
|----------------------------------------------|----------|
| Contact stomatitis | 10067510 |
| Contrast media allergy | 10066973 |
| Contrast media reaction | 10010836 |
| Corneal oedema | 10011033 |
| Cutaneous vasculitis | 10011686 |
| Dennie-Morgan fold | 10062918 |
| Dermatitis | 10012431 |
| Dermatitis acneiform | 10012432 |
| Dermatitis allergic | 10012434 |
| Dermatitis atopic | 10012438 |
| Dermatitis bullous | 10012441 |
| Dermatitis contact | 10012442 |
| Dermatitis exfoliative | 10012455 |
| Dermatitis exfoliative generalised | 10012456 |
| Dermatitis herpetiformis | 10012468 |
| Dermatitis infected | 10012470 |
| Dermatitis psoriasiform | 10058675 |
| Device allergy | 10072867 |
| Dialysis membrane reaction | 10076665 |
| Distributive shock | 10070559 |
| Documented hypersensitivity to administered | 10076470 |
| product | |
| Drug cross-reactivity | 10076743 |
| Drug eruption | 10013687 |
| Drug hypersensitivity | 10013700 |
| Drug provocation test | 10074350 |
| Drug reaction with eosinophilia and systemic | 10073508 |
| symptoms | |
| Eczema | 10014184 |
| Eczema infantile | 10014198 |
| Eczema nummular | 10014201 |
| Eczema vaccinatum | 10066042 |
| Eczema vesicular | 10058681 |
| Eczema weeping | 10055182 |
| Encephalitis allergic | 10056387 |
| Encephalopathy allergic | 10014627 |


| In 1 199 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | 10050115 |
|-----------------------------------------------|----------|
| Eosinophilic granulomatosis with polyangiitis | 10078117 |
| Epidermal necrosis | 10059284 |
| Epidermolysis | 10053177 |
| Epidermolysis bullosa | 10014989 |
| Epiglottic oedema | 10015029 |
| Erythema multiforme | 10015218 |
| Erythema nodosum | 10015226 |
| Exfoliative rash | 10064579 |
| Eye allergy | 10015907 |
| Eye oedema | 10052139 |
| Eye swelling | 10015967 |
| Eyelid oedema | 10015993 |
| Face oedema | 10016029 |
| Fixed eruption | 10016741 |
| Giant papillary conjunctivitis | 10018258 |
| Gingival oedema | 10049305 |
| Gingival swelling | 10018291 |
| Gleich's syndrome | 10066837 |
| Haemorrhagic urticaria | 10059499 |
| Hand dermatitis | 10058898 |
| Henoch-Schonlein purpura | 10019617 |
| Henoch-Schonlein purpura nephritis | 10069440 |
| Heparin-induced thrombocytopenia | 10062506 |
| Hereditary angioedema | 10019860 |
| Hypersensitivity | 10020751 |
| Hypersensitivity vasculitis | 10020764 |
| Idiopathic urticaria | 10021247 |
| Immediate post-injection reaction | 10067142 |
| Immune thrombocytopenic purpura | 10074667 |
| Immune tolerance induction | 10070581 |
| Immune-mediated adverse reaction | 10077665 |
| Implant site dermatitis | 10063855 |
| Implant site hypersensitivity | 10063858 |
| Implant site rash | 10063786 |
| Implant site urticaria | 10063787 |
| Incision site dermatitis | 10003787 |
| Interest of the defination | 100/3100 |


| | Incision site rash | 10073411 |
|---|---------------------------------------|----------|
| | Infusion site dermatitis | 10065458 |
| | Infusion site eczema | 10074850 |
| | Infusion site hypersensitivity | 10065471 |
| | Infusion site rash | 10059830 |
| | Infusion site recall reaction | 10076085 |
| | Infusion site urticaria | 10065490 |
| | Infusion site vasculitis | 10074851 |
| | Injection site dermatitis | 10022056 |
| | Injection site eczema | 10066221 |
| | Injection site hypersensitivity | 10022071 |
| | Injection site rash | 10022094 |
| | Injection site recall reaction | 10066797 |
| | Injection site urticaria | 10022107 |
| | Injection site vasculitis | 10067995 |
| | Instillation site hypersensitivity | 10073612 |
| | Instillation site rash | 10073622 |
| | Instillation site urticaria | 10073627 |
| | Interstitial granulomatous dermatitis | 10067972 |
| | Intestinal angioedema | 10076229 |
| | Iodine allergy | 10052098 |
| | Kaposi's varicelliform eruption | 10051891 |
| | Kounis syndrome | 10069167 |
| | Laryngeal oedema | 10023845 |
| | Laryngitis allergic | 10064866 |
| | Laryngospasm | 10023891 |
| | Laryngotracheal oedema | 10023893 |
| | Limbal swelling | 10070492 |
| | Lip oedema | 10024558 |
| | Lip swelling | 10024570 |
| | Mast cell degranulation present | 10076606 |
| | Medical device site dermatitis | 10075572 |
| | Medical device site eczema | 10075575 |
| | Medical device site hypersensitivity | 10075579 |
| | Medical device site rash | 10075585 |
| l | | |


| <br> | |
|-------------------------------------------------|----------|
| Medical device site urticaria | 10075588 |
| Mouth swelling | 10075203 |
| Mucocutaneous rash | 10056671 |
| Multiple allergies | 10028164 |
| Nephritis allergic | 10029120 |
| Nikolsky's sign | 10029415 |
| Nodular rash | 10075807 |
| Oculomucocutaneous syndrome | 10030081 |
| Oculorespiratory syndrome | 10067317 |
| Oedema mouth | 10030110 |
| Oral allergy syndrome | 10068355 |
| Oropharyngeal blistering | 10067950 |
| Oropharyngeal oedema | 10078783 |
| Oropharyngeal spasm | 10031111 |
| Oropharyngeal swelling | 10031118 |
| Palatal oedema | 10056998 |
| Palatal swelling | 10074403 |
| Palisaded neutrophilic granulomatous dermatitis | 10068809 |
| Palpable purpura | 10056872 |
| Pathergy reaction | 10074332 |
| Periorbital oedema | 10034545 |
| Pharyngeal oedema | 10034829 |
| Pruritus allergic | 10063438 |
| Radioallergosorbent test positive | 10037789 |
| Rash | 10037844 |
| Rash erythematous | 10037855 |
| Rash follicular | 10037857 |
| Rash generalised | 10037858 |
| Rash macular | 10037867 |
| Rash maculo-papular | 10037868 |
| Rash maculovesicular | 10050004 |
| Rash morbilliform | 10037870 |
| Rash neonatal | 10037871 |
| Rash papulosquamous | 10037879 |
| Rash pruritic | 10037884 |
| Rash pustular | 10037888 |
| 1 | 1 |


| Rash rubelliform | 10057984 |
|---------------------------------------------|----------|
| Rash scarlatiniform | 10037890 |
| Rash vesicular | 10037898 |
| Reaction to azo-dyes | 10037973 |
| Reaction to colouring | 10037974 |
| Reaction to drug excipients | 10064787 |
| Reaction to preservatives | 10064788 |
| Red man syndrome | 10038192 |
| Rhinitis allergic | 10039085 |
| Scleral oedema | 10057431 |
| Scleritis allergic | 10051126 |
| Scrotal oedema | 10039755 |
| Serum sickness | 10040400 |
| Serum sickness-like reaction | 10040402 |
| Shock | 10040560 |
| Shock symptom | 10040581 |
| Skin necrosis | 10040893 |
| Skin reaction | 10040914 |
| Skin test positive | 10040934 |
| Solar urticaria | 10041307 |
| Solvent sensitivity | 10041316 |
| Stevens-Johnson syndrome | 10042033 |
| Stoma site hypersensitivity | 10074509 |
| Stoma site rash | 10059071 |
| Swelling face | 10042682 |
| Swollen tongue | 10042727 |
| Symmetrical drug-related intertriginous and | 10078325 |
| flexural exanthema | |
| Tongue oedema | 10043967 |
| Toxic epidermal necrolysis | 10044223 |
| Toxic skin eruption | 10057970 |
| Tracheal oedema | 10044296 |
| Type I hypersensitivity | 10045240 |
| Type II hypersensitivity | 10054000 |
| Type III immune complex mediated reaction | 10053614 |
| Type IV hypersensitivity reaction | 10053613 |
| | 1 |


| Urticaria | 10046735 |
|-----------------------------------|----------|
| Urticaria cholinergic | 10046740 |
| Urticaria chronic | 10052568 |
| Urticaria contact | 10046742 |
| Urticaria papular | 10046750 |
| Urticaria physical | 10046751 |
| Urticaria pigmentosa | 10046752 |
| Urticaria vesiculosa | 10046755 |
| Urticarial vasculitis | 10048820 |
| Vaccination site dermatitis | 10069477 |
| Vaccination site eczema | 10076161 |
| Vaccination site exfoliation | 10069489 |
| Vaccination site hypersensitivity | 10068880 |
| Vaccination site rash | 10069482 |
| Vaccination site recall reaction | 10076188 |
| Vaccination site urticaria | 10069622 |
| Vaccination site vasculitis | 10076191 |
| Vaccination site vesicles | 10069623 |
| Vaginal exfoliation | 10064483 |
| Vaginal ulceration | 10046943 |
| Vasculitic rash | 10047111 |
| Vessel puncture site rash | 10077117 |
| Vessel puncture site vesicles | 10077813 |
| Vulval ulceration | 10047768 |
| Vulvovaginal rash | 10071588 |
| Vulvovaginal ulceration | 10050181 |


# 13.6.3 Bleeding Events

| ~ - | | PT | | | |
|---|---|---|---|---|---|
| Code | PT | Code | | | |
| 000039 | | 10067383<br>10067788 | | | |
| | | 10067788 | | | |
| | | 10058994 | | | |
| | | 10038994 | | | |
| | I | 10075094 | | | |
| | | 10075100 | | | |
| | | 10075100 | | | |
| | | 10059194 | | | |
| | _ | 10001361 | | | |
| | | 10049555 | | | |
| | | 10063896 | | | |
| | | 10056346 | | | |
| | | 10002244 | | | |
| | · · | 10048380 | | | |
| | | 10064223 | | | |
| | | 10068925 | | | |
| | | 10002886 | | | |
| | | 10068119 | | | |
| | Aortic intramural haematoma | 10067975 | | | |
| | Aortic perforation | 10075729 | | | |
| | Aortic rupture | 10060874 | | | |
| | Aponeurosis contusion | 10075330 | | | |
| | Application site bruise | 10050114 | | | |
| | | | İ | İ | Application site haematoma |
| | Application site haemorrhage | 10072694 | | | |
| | Application site purpura | 10050182 | | | |
| | Arterial haemorrhage | 10060964 | | | |
| | Arterial intramural haematoma | 10074971 | | | |
| | Arterial perforation | 10075732 | | | |
| | * | 10003173 | | | |
| | Arteriovenous fistula site haematoma | 10055150 | | | |
| | | 10055123 | | | |
| | _ | 10055152 | | | |
| | | 10055126 | | | |
| | 000039 | Abdominal wall haematoma Abdominal wall haemorrhage Abnormal withdrawal bleeding Acute haemorrhagic leukoencephalitis Acute haemorrhagic ulcerative colitis Administration site bruise Administration site haematoma Administration site haemorrhage Adrenal haematoma Adrenal haemorrhage Anal ulcer haemorrhage Anastomotic haemorrhage Anastomotic ulcer haemorrhage Aneurysm ruptured Angina bullosa haemorrhage Anorectal varices haemorrhage Aortic aneurysm rupture Aortic dissection rupture Aortic rupture Aortic rupture Aponeurosis contusion Application site bruise Application site haematoma Application site haemorrhage Arterial haemorrhage Arterial intramural haematoma Arterial perforation Arterial rupture | | | |


| MedDRA v20.0 | SMQ | | PT |
|--------------|------|------------------------------------|----------|
| SMQ | Code | PT | Code |
| | | Astringent therapy | 10067372 |
| | | Atrial rupture | 10048761 |
| | | Auricular haematoma | 10003797 |
| | | Basal ganglia haematoma | 10077031 |
| | | Basal ganglia haemorrhage | 10067057 |
| | | Basilar artery perforation | 10075736 |
| | | Bladder tamponade | 10062656 |
| | | Bleeding varicose vein | 10005144 |
| | | Blood blister | 10005372 |
| | | Blood urine | 10005863 |
| | | Blood urine present | 10018870 |
| | | Bloody discharge | 10057687 |
| | | Bloody peritoneal effluent | 10067442 |
| | | Bone contusion | 10066251 |
| | | Bone marrow haemorrhage | 10073581 |
| | | Brain contusion | 10052346 |
| | | Brain stem haematoma | 10073230 |
| | | Brain stem haemorrhage | 10006145 |
| | | Brain stem microhaemorrhage | 10071205 |
| | | Breast haematoma | 10064753 |
| | | Breast haemorrhage | 10006254 |
| | | Broad ligament haematoma | 10006375 |
| | | Bronchial haemorrhage | 10065739 |
| | | Bronchial varices haemorrhage | 10079163 |
| | | Bursal haematoma | 10077818 |
| | | Cardiac contusion | 10073356 |
| | | Carotid aneurysm rupture | 10051328 |
| | | Carotid artery perforation | 10075728 |
| | | Catheter site bruise | 10063587 |
| | | Catheter site haematoma | 10055662 |
| | | Catheter site haemorrhage | 10051099 |
| | | Central nervous system haemorrhage | 10072043 |
| | | Cephalhaematoma | 10008014 |
| | | Cerebellar haematoma | 10061038 |
| | | Cerebellar haemorrhage | 10008030 |
| | | Cerebellar microhaemorrhage | 10071206 |
| | | Cerebral aneurysm perforation | 10075394 |


| MedDRA v20.0 | SMQ | | PT |
|---|---|---|---|
| SMQ | Code | PT | Code |
| | | Cerebral aneurysm ruptured syphilitic | 10008076 |
| | | Cerebral arteriovenous malformation haemorrhagic | 10008086 |
| | | Cerebral artery perforation | 10075734 |
| | | Cerebral haematoma | 10053942 |
| | | Cerebral haemorrhage | 10008111 |
| | | Cerebral haemorrhage foetal | 10050157 |
| | | Cerebral haemorrhage neonatal | 10008112 |
| | | Cerebral microhaemorrhage | 10067277 |
| | | Cervix haematoma uterine | 10050020 |
| | | Cervix haemorrhage uterine | 10050022 |
| | | Chest wall haematoma | 10076597 |
| | | Choroidal haematoma | 10068642 |
| | | Choroidal haemorrhage | 10008786 |
| | | Chronic gastrointestinal bleeding | 10050399 |
| | | Chronic pigmented purpura | 10072726 |
| | | Ciliary body haemorrhage | 10057417 |
| | | Coital bleeding | 10065019 |
| | | Colonic haematoma | 10009996 |
| | | Conjunctival haemorrhage | 10010719 |
| | | Contusion | 10050584 |
| | | Corneal bleeding | 10051558 |
| | | Cullen's sign | 10059029 |
| | | Cystitis haemorrhagic | 10011793 |
| | | Deep dissecting haematoma | 10074718 |
| | | Diarrhoea haemorrhagic | 10012741 |
| | | Disseminated intravascular coagulation | 10013442 |
| | | Diverticulitis intestinal haemorrhagic | 10013541 |
| | | Diverticulum intestinal haemorrhagic | 10013560 |
| | | Duodenal ulcer haemorrhage | 10013839 |
| | | Duodenitis haemorrhagic | 10013865 |
| | | Dysfunctional uterine bleeding | 10013908 |
| | | Ear haemorrhage | 10014009 |
| | | Ecchymosis | 10014080 |
| | | Encephalitis haemorrhagic | 10014589 |
| | | Enterocolitis haemorrhagic | 10014896 |
| | | Epidural haemorrhage | 10073681 |
| | | Epistaxis | 10015090 |


| MedDRA v20.0 | SMQ | | PT |
|---|---|---|---|
| SMQ | Code | PT | Code |
| | | Exsanguination | 10015719 |
| | | Extra-axial haemorrhage | 10078254 |
| | | Extradural haematoma | 10015769 |
| | | Extravasation blood | 10015867 |
| | | Eye contusion | 10073354 |
| | | Eye haemorrhage | 10015926 |
| | | Eyelid bleeding | 10053196 |
| | | Eyelid contusion | 10075018 |
| | | Eyelid haematoma | 10064976 |
| | | Femoral artery perforation | 10075739 |
| | | Femoral vein perforation | 10075745 |
| | | Foetal-maternal haemorrhage | 10016871 |
| | | Gastric haemorrhage | 10017788 |
| | | Gastric ulcer haemorrhage | 10017826 |
| | | Gastric ulcer haemorrhage, obstructive | 10017829 |
| | | Gastric varices haemorrhage | 10057572 |
| | | Gastritis alcoholic haemorrhagic | 10017857 |
| | | Gastritis haemorrhagic | 10017866 |
| | | Gastroduodenal haemorrhage | 10053768 |
| | | Gastroduodenitis haemorrhagic | 10048712 |
| | | Gastrointestinal angiodysplasia haemorrhagic | 10017929 |
| | | Gastrointestinal haemorrhage | 10017955 |
| | | Gastrointestinal polyp haemorrhage | 10074437 |
| | | Gastrointestinal ulcer haemorrhage | 10056743 |
| | | Genital contusion | 10073355 |
| | | Genital haemorrhage | 10061178 |
| | | Gingival bleeding | 10018276 |
| | | Graft haemorrhage | 10063577 |
| | | Grey Turner's sign | 10075426 |
| | | Haemarthrosis | 10018829 |
| | | Haematemesis | 10018830 |
| | | Haematochezia | 10018836 |
| | | Haematocoele | 10018833 |
| | | Haematoma | 10018852 |
| | | Haematoma evacuation | 10060733 |
| | | Haematoma infection | 10051564 |
| | | Haematosalpinx | 10050468 |


| MedDRA v20.0 | SMQ | | PT |
|--------------|------|-----------------------------------------|----------|
| SMQ | Code | PT | Code |
| | | Haematospermia | 10018866 |
| | | Haematotympanum | 10063013 |
| | | Haematuria | 10018867 |
| | | Haematuria traumatic | 10018871 |
| | | Haemobilia | 10058947 |
| | | Haemophilic arthropathy | 10065057 |
| | | Haemoptysis | 10018964 |
| | | Haemorrhage | 10055798 |
| | | Haemorrhage coronary artery | 10055803 |
| | | Haemorrhage foetal | 10061191 |
| | | Haemorrhage in pregnancy | 10018981 |
| | | Haemorrhage intracranial | 10018985 |
| | | Haemorrhage neonatal | 10061993 |
| | | Haemorrhage subcutaneous | 10018999 |
| | | Haemorrhage subepidermal | 10019001 |
| | | Haemorrhage urinary tract | 10055847 |
| | | Haemorrhagic anaemia | 10052293 |
| | | Haemorrhagic arteriovenous malformation | 10064595 |
| | | Haemorrhagic ascites | 10059766 |
| | | Haemorrhagic breast cyst | 10077443 |
| | | Haemorrhagic cerebral infarction | 10019005 |
| | | Haemorrhagic cyst | 10059189 |
| | | Haemorrhagic diathesis | 10062713 |
| | | Haemorrhagic disease of newborn | 10019008 |
| | | Haemorrhagic disorder | 10019009 |
| | | Haemorrhagic erosive gastritis | 10067786 |
| | | Haemorrhagic hepatic cyst | 10067796 |
| | | Haemorrhagic infarction | 10019013 |
| | | Haemorrhagic necrotic pancreatitis | 10076058 |
| | | Haemorrhagic ovarian cyst | 10060781 |
| | | Haemorrhagic stroke | 10019016 |
| | | Haemorrhagic thyroid cyst | 10072256 |
| | | Haemorrhagic transformation stroke | 10055677 |
| | | Haemorrhagic tumour necrosis | 10054096 |
| | | Haemorrhagic urticaria | 10059499 |
| | | Haemorrhagic vasculitis | 10071252 |
| | | Haemorrhoidal haemorrhage | 10054787 |


| MedDRA v20.0 | SMQ | | PT |
|--------------|------|----------------------------------------|----------|
| SMQ | Code | PT | Code |
| | | Haemostasis | 10067439 |
| | | Haemothorax | 10019027 |
| | | Henoch-Schonlein purpura | 10019617 |
| | | Hepatic haemangioma rupture | 10054885 |
| | | Hepatic haematoma | 10019676 |
| | | Hepatic haemorrhage | 10019677 |
| | | Hereditary haemorrhagic telangiectasia | 10019883 |
| | | Hyperfibrinolysis | 10074737 |
| | | Hyphaema | 10020923 |
| | | Iliac artery perforation | 10075731 |
| | | Iliac artery rupture | 10072789 |
| | | Iliac vein perforation | 10075744 |
| | | Immune thrombocytopenic purpura | 10074667 |
| | | Implant site bruising | 10063850 |
| | | Implant site haematoma | 10063780 |
| | | Implant site haemorrhage | 10053995 |
| | | Incision site haematoma | 10059241 |
| | | Incision site haemorrhage | 10051100 |
| | | Increased tendency to bruise | 10021688 |
| | | Induced abortion haemorrhage | 10052844 |
| | | Inferior vena cava perforation | 10075742 |
| | | Infusion site bruising | 10059203 |
| | | Infusion site haematoma | 10065463 |
| | | Infusion site haemorrhage | 10065464 |
| | | Injection site bruising | 10022052 |
| | | Injection site haematoma | 10022066 |
| | | Injection site haemorrhage | 10022067 |
| | | Instillation site bruise | 10073630 |
| | | Instillation site haematoma | 10073609 |
| | | Instillation site haemorrhage | 10073610 |
| | | Internal haemorrhage | 10075192 |
| | | Intestinal haematoma | 10069829 |
| | | Intestinal haemorrhage | 10059175 |
| | | Intestinal varices haemorrhage | 10078058 |
| | | Intra-abdominal haematoma | 10056457 |
| | | Intra-abdominal haemorrhage | 10061249 |
| | | Intracerebral haematoma evacuation | 10062025 |


| MedDRA v20.0 | SMQ | | PT |
|--------------|------|---------------------------------------|----------|
| SMQ | Code | PT | Code |
| | | Intracranial haematoma | 10059491 |
| | | Intracranial tumour haemorrhage | 10022775 |
| | | Intraocular haematoma | 10071934 |
| | | Intrapartum haemorrhage | 10067703 |
| | | Intraventricular haemorrhage | 10022840 |
| | | Intraventricular haemorrhage neonatal | 10022841 |
| | | Iris haemorrhage | 10057418 |
| | | Joint microhaemorrhage | 10077666 |
| | | Kidney contusion | 10023413 |
| | | Lacrimal haemorrhage | 10069930 |
| | | Large intestinal haemorrhage | 10052534 |
| | | Large intestinal ulcer haemorrhage | 10061262 |
| | | Laryngeal haematoma | 10070885 |
| | | Laryngeal haemorrhage | 10065740 |
| | | Lip haematoma | 10066304 |
| | | Lip haemorrhage | 10049297 |
| | | Liver contusion | 10067266 |
| | | Lower gastrointestinal haemorrhage | 10050953 |
| | | Lower limb artery perforation | 10075730 |
| | | Lymph node haemorrhage | 10074270 |
| | | Mallory-Weiss syndrome | 10026712 |
| | | Mediastinal haematoma | 10049941 |
| | | Mediastinal haemorrhage | 10056343 |
| | | Medical device site bruise | 10075570 |
| | | Medical device site haematoma | 10075577 |
| | | Medical device site haemorrhage | 10075578 |
| | | Melaena | 10027141 |
| | | Melaena neonatal | 10049777 |
| | | Meningorrhagia | 10052593 |
| | | Menometrorrhagia | 10027295 |
| | | Menorrhagia | 10027313 |
| | | Mesenteric haematoma | 10071557 |
| | | Mesenteric haemorrhage | 10060717 |
| | | Metrorrhagia | 10027514 |
| | | Mouth haemorrhage | 10028024 |
| | | Mucocutaneous haemorrhage | 10076048 |
| | | Mucosal haemorrhage | 10061298 |


| MedDRA v20.0 | SMQ | | PT |
|--------------|------|---------------------------------------|----------|
| SMQ | Code | PT | Code |
| | | Muscle contusion | 10070757 |
| | | Muscle haemorrhage | 10028309 |
| | | Myocardial haemorrhage | 10048849 |
| | | Myocardial rupture | 10028604 |
| | | Naevus haemorrhage | 10062955 |
| | | Nail bed bleeding | 10048891 |
| | | Nasal septum haematoma | 10075027 |
| | | Neonatal gastrointestinal haemorrhage | 10074159 |
| | | Nephritis haemorrhagic | 10029132 |
| | | Nipple exudate bloody | 10029418 |
| | | Ocular retrobulbar haemorrhage | 10057571 |
| | | Oesophageal haemorrhage | 10030172 |
| | | Oesophageal intramural haematoma | 10077486 |
| | | Oesophageal ulcer haemorrhage | 10030202 |
| | | Oesophageal varices haemorrhage | 10030210 |
| | | Oesophagitis haemorrhagic | 10030219 |
| | | Optic disc haemorrhage | 10030919 |
| | | Optic nerve sheath haemorrhage | 10030941 |
| | | Oral contusion | 10078170 |
| | | Oral mucosa haematoma | 10074779 |
| | | Osteorrhagia | 10051937 |
| | | Ovarian haematoma | 10033263 |
| | | Ovarian haemorrhage | 10065741 |
| | | Palpable purpura | 10056872 |
| | | Pancreatic haemorrhage | 10033625 |
| | | Pancreatitis haemorrhagic | 10033650 |
| | | Papillary muscle haemorrhage | 10059164 |
| | | Paranasal sinus haematoma | 10069702 |
| | | Parathyroid haemorrhage | 10059051 |
| | | Parotid gland haemorrhage | 10051166 |
| | | Pelvic haematoma | 10054974 |
| | | Pelvic haematoma obstetric | 10034248 |
| | | Pelvic haemorrhage | 10063678 |
| | | Penile contusion | 10073352 |
| | | Penile haematoma | 10070656 |
| | | Penile haemorrhage | 10034305 |
| | | Peptic ulcer haemorrhage | 10034344 |


| MedDRA v20.0 | SMQ | | PT |
|---|---|---|---|
| SMQ | Code | PT | Code |
| | | Pericardial haemorrhage | 10034476 |
| | | Perineal haematoma | 10034520 |
| | | Periorbital haematoma | 10034544 |
| | | Periorbital haemorrhage | 10071697 |
| | | Periosteal haematoma | 10077341 |
| | | Peripartum haemorrhage | 10072693 |
| | | Perirenal haematoma | 10049450 |
| | | Peritoneal haematoma | 10058095 |
| | | Peritoneal haemorrhage | 10034666 |
| | | Periventricular haemorrhage neonatal | 10076706 |
| | | Petechiae | 10034754 |
| | | Pharyngeal haematoma | 10068121 |
| | | Pharyngeal haemorrhage | 10034827 |
| | | Pituitary haemorrhage | 10049760 |
| | | Placenta praevia haemorrhage | 10035121 |
| | | Polymenorrhagia | 10064050 |
| | | Post abortion haemorrhage | 10036246 |
| | | Post procedural contusion | 10073353 |
| | | Post procedural haematoma | 10063188 |
| | | Post procedural haematuria | 10066225 |
| | | Post procedural haemorrhage | 10051077 |
| | | Post transfusion purpura | 10072265 |
| | | Postmenopausal haemorrhage | 10055870 |
| | | Postpartum haemorrhage | 10036417 |
| | | Post-traumatic punctate intraepidermal haemorrhage | 10071639 |
| | | Premature separation of placenta | 10036608 |
| | | Procedural haemorrhage | 10071229 |
| | | Proctitis haemorrhagic | 10036778 |
| | | Prostatic haemorrhage | 10036960 |
| | | Pulmonary alveolar haemorrhage | 10037313 |
| | | Pulmonary contusion | 10037370 |
| | | Pulmonary haematoma | 10054991 |
| | | Pulmonary haemorrhage | 10037394 |
| | | Puncture site haemorrhage | 10051101 |
| | | Purpura | 10037549 |
| | | Purpura fulminans | 10037556 |
| | | Purpura neonatal | 10037557 |


| MedDRA v20.0 | SMQ | | PT |
|--------------|------|----------------------------------------|----------|
| SMQ | Code | PT | Code |
| | | Purpura non-thrombocytopenic | 10057739 |
| | | Purpura senile | 10037560 |
| | | Putamen haemorrhage | 10058940 |
| | | Radiation associated haemorrhage | 10072281 |
| | | Rectal haemorrhage | 10038063 |
| | | Rectal ulcer haemorrhage | 10038081 |
| | | Renal artery perforation | 10075737 |
| | | Renal cyst haemorrhage | 10059846 |
| | | Renal haematoma | 10038459 |
| | | Renal haemorrhage | 10038460 |
| | | Respiratory tract haemorrhage | 10038727 |
| | | Respiratory tract haemorrhage neonatal | 10038728 |
| | | Retinal aneurysm rupture | 10079121 |
| | | Retinal haemorrhage | 10038867 |
| | | Retinopathy haemorrhagic | 10051447 |
| | | Retroperitoneal haematoma | 10058360 |
| | | Retroperitoneal haemorrhage | 10038980 |
| | | Retroplacental haematoma | 10054798 |
| | | Ruptured cerebral aneurysm | 10039330 |
| | | Scleral haemorrhage | 10050508 |
| | | Scrotal haematocoele | 10061517 |
| | | Scrotal haematoma | 10039749 |
| | | Shock haemorrhagic | 10049771 |
| | | Skin haemorrhage | 10064265 |
| | | Skin neoplasm bleeding | 10060712 |
| | | Skin ulcer haemorrhage | 10050377 |
| | | Small intestinal haemorrhage | 10052535 |
| | | Small intestinal ulcer haemorrhage | 10061550 |
| | | Soft tissue haemorrhage | 10051297 |
| | | Spermatic cord haemorrhage | 10065742 |
| | | Spinal cord haematoma | 10076051 |
| | | Spinal cord haemorrhage | 10048992 |
| | | Spinal epidural haematoma | 10050162 |
| | | Spinal epidural haemorrhage | 10049236 |
| | | Spinal subarachnoid haemorrhage | 10073564 |
| | | Spinal subdural haematoma | 10050164 |
| | | Spinal subdural haemorrhage | 10073563 |


| MedDRA v20.0 | SMQ | | PT |
|--------------|------|-------------------------------------|----------|
| SMQ | Code | PT | Code |
| | | Spleen contusion | 10073533 |
| | | Splenic artery perforation | 10075738 |
| | | Splenic haematoma | 10041646 |
| | | Splenic haemorrhage | 10041647 |
| | | Splenic varices haemorrhage | 10068662 |
| | | Splinter haemorrhages | 10041663 |
| | | Spontaneous haematoma | 10065304 |
| | | Spontaneous haemorrhage | 10074557 |
| | | Stoma site haemorrhage | 10074508 |
| | | Stomatitis haemorrhagic | 10042132 |
| | | Subarachnoid haematoma | 10076701 |
| | | Subarachnoid haemorrhage | 10042316 |
| | | Subarachnoid haemorrhage neonatal | 10042317 |
| | | Subchorionic haematoma | 10072596 |
| | | Subchorionic haemorrhage | 10071010 |
| | | Subclavian artery perforation | 10075740 |
| | | Subclavian vein perforation | 10075743 |
| | | Subcutaneous haematoma | 10042345 |
| | | Subdural haematoma | 10042361 |
| | | Subdural haematoma evacuation | 10042363 |
| | | Subdural haemorrhage | 10042364 |
| | | Subdural haemorrhage neonatal | 10042365 |
| | | Subgaleal haematoma | 10069510 |
| | | Subretinal haematoma | 10071935 |
| | | Superior vena cava perforation | 10075741 |
| | | Testicular haemorrhage | 10051877 |
| | | Thalamus haemorrhage | 10058939 |
| | | Third stage postpartum haemorrhage | 10043449 |
| | | Thoracic haemorrhage | 10062744 |
| | | Thrombocytopenic purpura | 10043561 |
| | | Thrombotic thrombocytopenic purpura | 10043648 |
| | | Thyroid haemorrhage | 10064224 |
| | | Tongue haematoma | 10043959 |
| | | Tongue haemorrhage | 10049870 |
| | | Tonsillar haemorrhage | 10057450 |
| | | Tooth pulp haemorrhage | 10072228 |
| | | Tooth socket haemorrhage | 10064946 |


| MedDRA v20.0 | SMQ | | PT |
|--------------|------|------------------------------------|----------|
| SMQ | Code | PT | Code |
| | | Tracheal haemorrhage | 10062543 |
| | | Traumatic haematoma | 10044522 |
| | | Traumatic haemorrhage | 10053476 |
| | | Traumatic haemothorax | 10074487 |
| | | Traumatic intracranial haematoma | 10079013 |
| | | Traumatic intracranial haemorrhage | 10061387 |
| | | Tumour haemorrhage | 10049750 |
| | | Ulcer haemorrhage | 10061577 |
| | | Umbilical cord haemorrhage | 10064534 |
| | | Umbilical haematoma | 10068712 |
| | | Umbilical haemorrhage | 10045455 |
| | | Upper gastrointestinal haemorrhage | 10046274 |
| | | Ureteric haemorrhage | 10065743 |
| | | Urethral haemorrhage | 10049710 |
| | | Urinary bladder haemorrhage | 10046528 |
| | | Urogenital haemorrhage | 10050058 |
| | | Uterine haematoma | 10063875 |
| | | Uterine haemorrhage | 10046788 |
| | | Vaccination site bruising | 10069484 |
| | | Vaccination site haematoma | 10069472 |
| | | Vaccination site haemorrhage | 10069475 |
| | | Vaginal haematoma | 10046909 |
| | | Vaginal haemorrhage | 10046910 |
| | | Varicose vein ruptured | 10046999 |
| | | Vascular access site bruising | 10077767 |
| | | Vascular access site haematoma | 10077647 |
| | | Vascular access site haemorrhage | 10077643 |
| | | Vascular access site rupture | 10077652 |
| | | Vascular graft haemorrhage | 10077721 |
| | | Vascular pseudoaneurysm ruptured | 10053949 |
| | | Vascular purpura | 10047097 |
| | | Vascular rupture | 10053649 |
| | | Vein rupture | 10077110 |
| | | Venous haemorrhage | 10065441 |
| | | Venous perforation | 10075733 |
| | | Ventricle rupture | 10047279 |
| | | Vertebral artery perforation | 10075735 |


Statistical Analysis Plan

Protocol Number: CSL112\_2001 Product Name: CSL112

| MedDRA v20.0<br>SMQ | SMQ<br>Code | PT | PT<br>Code |
|---|---|---|---|
| | | Vessel puncture site bruise | 10063881 |
| | | Vessel puncture site haematoma | 10065902 |
| | | Vessel puncture site haemorrhage | 10054092 |
| | | Vitreous haematoma | 10071936 |
| | | Vitreous haemorrhage | 10047655 |
| | | Vulval haematoma | 10047756 |
| | | Vulval haematoma evacuation | 10047757 |
| | | Vulval haemorrhage | 10063816 |
| | | Withdrawal bleed | 10047998 |
| | | Wound haematoma | 10071504 |
| | | Wound haemorrhage | 10051373 |


# 13.6.4 Hemolysis

| MedDRA v20.0<br>SMQ | SMQ<br>Code | PT | PT<br>Code |
|---|---|---|---|
| Haemolytic | 20000019 | ABO haemolytic disease of newborn | 10000205 |
| Disorders, Narrow | | ABO incompatibility | 10000206 |
| | | Acid haemolysin test positive | 10073783 |
| | | Acute haemolytic transfusion reaction | 10066181 |
| | | Alloimmunisation | 10060935 |
| | | Anti A antibody positive | 10074302 |
| | | Anti B antibody positive | 10074303 |
| | | Anti Kell antibody test positive | 10078305 |
| | | Anti-erythrocyte antibody positive | 10057108 |
| | | Autoimmune haemolytic anaemia | 10073785 |
| | | Blood incompatibility haemolytic anaemia of newborn | 10056369 |
| | | Cardiac haemolytic anaemia | 10072202 |
| | | Cold agglutinins positive | 10009854 |
| | | Cold type haemolytic anaemia | 10009868 |
| | | Coombs direct test positive | 10010933 |
| | | Coombs indirect test positive | 10010938 |
| | | Coombs negative haemolytic anaemia | 10010940 |
| | | Coombs positive haemolytic anaemia | 10010941 |
| | | Coombs test positive | 10061090 |
| | | Delayed haemolytic transfusion reaction | 10066182 |
| | | Erythroblastosis | 10049466 |
| | | Erythroblastosis foetalis | 10015251 |
| | | Evans syndrome | 10053873 |
| | | Extravascular haemolysis | 10015871 |
| | | Glucose-6-phosphate dehydrogenase abnormal | 10059902 |
| | | Glucose-6-phosphate dehydrogenase deficiency | 10018444 |
| | | Haemoglobin urine present | 10018909 |
| | | Haemoglobinaemia | 10018901 |
| | | Haemoglobinuria | 10018906 |
| | | Haemolysis | 10018910 |
| | | Haemolysis neonatal | 10050190 |
| | | Haemolytic anaemia | 10018916 |
| | | Haemolytic transfusion reaction | 10067122 |
| | | Haemolytic uraemic syndrome | 10018932 |
| | | Haemosiderinuria | 10069395 |


| Г | | |
|---|--------------------------------------|----------|
| | Haptoglobin decreased | 10019150 |
| | Intravascular haemolysis | 10022822 |
| | Isoimmune haemolytic disease | 10023052 |
| | Jaundice acholuric | 10023128 |
| | Microangiopathic haemolytic anaemia | 10027527 |
| | Paroxysmal nocturnal haemoglobinuria | 10034042 |
| | Passenger lymphocyte syndrome | 10073596 |
| | Red cell fragmentation syndrome | 10072203 |
| | Rhesus antibodies positive | 10039036 |
| | Rhesus haemolytic disease of newborn | 10039037 |
| | Rhesus incompatibility | 10063676 |
| | Schistocytosis | 10076534 |
| | Transfusion reaction | 10044359 |
| | Warm type haemolytic anaemia | 10047822 |

# 13.7 Source Data for Identifying Baseline Medications of Interest

CSLCT-HDL-12-77\_w hodrug\_unqiue\_28Ju


# Signature Page

CSL112\_2001 - Statistical Analysis Plan - v1 - 03Aug2017

| Signed By Date (GMT) |
|----------------------|
|----------------------|

Signature Page 1 of 1

--- Do Not Detach This Signature Page ---

glbdctmp Print Date: 21-Jan-2020 08:18:18 GMT-05:00